Title: A Randomized, Phase II Study of Ficlatuzumab with or without Cetuximab in Patients with Cetuximab-Resistant, Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma



**UA IRB Protocol #:** 1710965268

**IND#:** 136947 (Research IND)

Phase: II Version: V. 10

Investigational Agent: Ficlatuzumab
Commercial Agent: Cetuximab

#### **CO-PRINICPAL INVESTIGATOR:**

Ricklie Julian, MD

University of Arizona Cancer Center

1515 N. Campbell Ave. Tucson, AZ 85724 Phone: 520-694-2873 Email: rickliej@arizona.edu

#### **CO-PRINICPAL INVESTIGATOR & SPONSOR-INVESTIGATOR:**

Julie E. Bauman, MD, MPH

University of Arizona Cancer Center

1515 N. Campbell Ave. Tucson, AZ 85724

Email: jebauman@email.arizona.edu

**Source(s) of Support**: Aveo Oncology

Aveo Oncology Protocol ID #: AV-299-17-117i

**Study Safety Oversight**: University of Arizona Cancer Center

Data Safety and Monitoring Board

 v10, 05/23/2023

## **TRIAL SCHEMA**



# TABLE OF CONTENTS

| 1. | BACKGROUND & RATIONA | \LE | 6 |
|---|---|---|---|
| 1.1 | | | |
| 1.2 | | eceptor in HNSCC | |
| 1.3 | | eck Squamous Cell Carcinoma | |
| 1.4 | • | oination of Ficlatuzumab and Cetuximab | |
| 1.5 | • | | |
| 1.6 | , , | | |
| | | xperience | |
| . <b>.</b> | · | perience | |
| 1.7 | | | |
| | | CC | |
| | | Week Dosing Schedule of Cetuximab | |
| 1.8 | Correlative Studies Backgro | ound | 15 |
| | 1.8.1 Tumoral Activation of H | HGF/cMet Pathway | 15 |
| | • | of HGF/cMet Pathway Activation | |
| | | IK3CA, PTEN, and HRAS | |
| | ' | omes | |
| 2. | STUDY OBJECTIVES | | 18 |
| 2.1 | Primary | | 18 |
| 2.2 | | | |
| 2.3 | Exploratory | | 18 |
| 3. | PATIENT SELECTION | | 18 |
| 3.1 | Inclusion Criteria | | 18 |
| 3.2 | Exclusion Criteria | | 21 |
| 4. | PATIENT REGISTRATION A | ND RANDOMIZATION | 23 |
| 4.1 | Registration | | 23 |
| 4.2 | 3 | | |
| 5. | TREATMENT PLAN | | 24 |
| 5.1 | | | |
| 5.1 | | n | |
| | | n for Arm B (Combination Arm) | |
| 5.2 | | | |
| ٥.۷ | | | |
| | | n | |
| | | n for Arm B (Combination Arm) | |
| | | TIOFATTI B (COMBINATION ATTI) | |
| 5.3 | | cation and Supportive Care Guidelines | |
| J.S | General Conconnitant Medi | caudii ailu suppoitive cale Guluelliles | ∠0 |

| 5.4 | Du | ration of Treatment and Follow-up | 26 |
|---|---|---|---|
| | 5.4.1 | Treatment Duration: | 26 |
| | 5.4.2 | Follow up duration - WITHOUT progressive disease: | 26 |
| | 5.4.3 | Follow up duration - WITH progressive disease: | |
| | 5.4.4 | Follow up for unacceptable adverse events | |
| 5.5 | Do | se Delays and Modifications | 27 |
| | 5.5.1 | Treatment Plan Interruptions and Delays | 27 |
| | 5.5.2 | Dose Reduction Levels | |
| | 5.5.3 | Treatment Stoppage Rules For Toxicity | |
| | 5.5.4 | Treatment Interruption for Interstitial Lung Disease | 28 |
| | 5.5.5 | Dose Modification for Hematologic Toxicity | 28 |
| | 5.5.6 | Dose Modification for Non-Hematologic Toxicity | 29 |
| | 5.5.7 | Dermatologic Toxicity | 35 |
| | 5.5.8 | Cetuximab Infusion Reaction | 37 |
| 6. | RES | SPONSE ASSESSMENT | 39 |
| 6.1 | Ма | lignant Disease Evaluation | 39 |
| | 6.1.1 | Measurable Disease | 40 |
| | 6.1.2 | Non-measurable disease | 40 |
| | 6.1.3 | Target Lesions | 40 |
| | 6.1.4 | Non-target Lesions | 41 |
| 6.2 | Res | sponse Criteria | 41 |
| | 6.2.1 | Evaluation of Target Lesions | 41 |
| | 6.2.2 | Evaluation of Non-target Lesions | 41 |
| | 6.2.3 | Evaluation of Patient's Best Overall Response | 42 |
| 6.3 | Ме | thods of Measurement | 44 |
| 7. | DR | UG INFORMATION | 46 |
| 7.1 | Fic | atuzumab | 46 |
| | 7.1.1 | Study Drug Materials | 46 |
| | 7.1.2 | Ficlatuzumab Study Drug Storage | |
| | 7.1.3 | Study Drug Accountability | |
| 7.2 | Cet | tuximab | |
| 8. | STU | JDY PROCEDURES/EVALUATIONS | 49 |
| 8.1 | Scr | eening/Pre-treatment evaluations | 49 |
| 8.2 | | gistration & Randomization | |
| 8.3 | | sluations during study treatment | |
| | 8.3.1 | Every Two Weeks – Day 1 and Day 15 of each cycle (+/- 3 days) | |
| | 8.3.2 | Every 8 Weeks (the end of even cycles – "Day 28"/8 weeks, 16 weeks, etc.) | |
| | 8.3.3 | OPTIONAL: Every 12 Weeks Cycle 13+ ("Day 28" of every 3 <sup>rd</sup> cycle after Cycle 12) | |
| 8.4 | Fno | d-of-treatment (EOT) evaluations | |
| 8.5 | | st-treatment follow-up | |
| 5 | 8.5.1 | Adverse Event and Concomitant Medication Follow-up | |
| | 8.5.2 | Discontinuation of treatment WITHOUT progressive disease | |

| 8. | 5.3 Progressive disease follow-up | 55 |
|---|---|---|
| 9. | BIOMARKER, CORRELATIVE, OR SPECIAL STUDIES | 55 |
| 9.1 | Submission of archived diagnostic tissue | 55 |
| 9.2 | Research biopsy | 55 |
| 9. | 2.1 Research Biopsy Methodology | 56 |
| 9.3 | Research Blood | 56 |
| 10. | STATISTICAL METHODS | 56 |
| 10.1 | Study Design | 56 |
| 10.2 | Primary Objective | |
| 10.3 | Sample Size Determination | |
| 10.4 | Secondary Objectives | 57 |
| | 0.4.1 Toxicity | |
| 10 | 0.4.2 Other Efficacy Endpoints | |
| 10.5 | Exploratory Objectives | 58 |
| | 0.5.1 Patient-Reported Outcomes | |
| 10 | 0.5.2 Biomarker endpoints | 58 |
| 10.6 | Statistical Analysis Plan | |
| 10.7 | Continuous Monitoring Rule for Futility | 58 |
| 11. | DATA SAFETY MONITORING PLAN | 59 |
| 12. | ADVERSE EVENT REPORTING | 62 |
| 12.1 | Definitions | 62 |
| 12.2 | Description of Adverse Event Reporting Procedures | |
| 12.3 | Reporting of Serious Adverse Events | |
| 12.4 | Review of Safety Information: Sponsor-Investigator Responsibilities | |
| 12.5 | IND safety reports for ficlatuzumab | |
| 13. | DATA HANDLING AND RECORD-KEEPING | |
| 14. | ETHICS AND REGULATORY COMPLIANCE | |
| 14.1 | Institutional Review Board (IRB) approval | |
| 14.2 | Ethical and scientific conduct of the clinical research study | |
| 14.3<br>14.4 | Subject informed consent | |
| | • | |
| | Cetux Protocol Signature Page | |
| 15. | APPENDICES | |
| 15.1 | Appendix A: FACT-H&N Symptom index (FHNSI) | |
| 15.2<br>15.3 | Appendix G: Study Calandar (Alca see Section 8) | |
| 15.3 | Appendix C: Study Calendar (Also see Section 8) | |
| 16. | REFERENCES | |
| 10. | NLI LNLINCE) | <i>1</i> 4 |

#### 1. BACKGROUND & RATIONALE

### 1.1 Background

Head and neck squamous cell carcinoma (HNSCC) is the most common cancer arising in the upper aerodigestive tract. HNSCC is the sixth leading incident cancer worldwide with 600,000 cases anticipated in 2012.<sup>1</sup> Despite advances in multimodality therapy, 5-year overall survival (OS) is 40-50%, and has increased only incrementally in the past two decades.<sup>2</sup> Patients with recurrent or metastatic (R/M) HNSCC have particularly poor prognosis, with median overall survival of 6-10 months. Options for palliative management are limited. For nearly three decades, the cornerstone of first line chemotherapy has been cisplatin,<sup>3</sup> frequently combined with fluorouracil or a taxane derivative due to increased response rate (RR) albeit no conclusive evidence of superior survival compared to cisplatin monotherapy.<sup>4</sup>

Ubiquitous expression of EGFR compelled the development of EGFR inhibitors for HNSCC treatment <sup>5, 6</sup>. The EGFR-directed monoclonal antibody, cetuximab, is the only targeted therapy to date FDA-approved for the treatment of HNSCC, and improves survival when added to front line platinum <sup>7</sup>. Despite aberrant EGFR signaling in the majority of HNSCC cases, the modest clinical activity of cetuximab has been disappointing; either primary or acquired resistance is inevitable. Co-targeting EGFR and a parallel or compensatory oncogenic pathway may overcome cetuximab resistance.

While immunotherapeutic antibodies inhibiting programmed death receptor 1 (PD-1) recently gained FDA approval in patients with platinum-refractory HNSCC, the OS benefit appears to be limited to approximately 20% <sup>8, 9</sup>. Currently, there is no standard therapy for patients after failure of platinum, cetuximab, and anti-PD1 therapy; all such patients will succumb with a median survival of less than 6 months. The lack of therapeutic options for patients with pan-refractory, recurrent and/or metastatic HNSCC represents a major unmet clinical need.

## 1.2 Epidermal Growth Factor Receptor in HNSCC

EGFR is a member of the ErbB/HER family of transmembrane glycoprotein receptor tyrosine kinases (RTK). Activated EGFR initiates a pleiotropic network of downstream signaling cascades including Ras/Raf/MAPK, PI3K/Akt, STAT, and Src Kinase effecting cellular proliferation, invasion, angiogenesis and metastasis. <sup>10</sup> *In vitro*, forced overexpression of EGFR causes malignant transformation of oral epithelial cells, suggesting its role as an oncogene in HNSCC. EGFR overexpression as measured by immunohistochemistry (IHC) and increased EGFR gene copy number as measured by fluorescence in situ hybridization occur in the majority of HNSCC, and associate with increased stage as well as reduced relapse-free and overall survival (OS). <sup>6, 11-13</sup> Thus, EGFR is both oncogene and prognostic biomarker in HNSCC.

EGFR's functional importance in HNSCC resulted in successful development of the first molecularly targeted strategy, the murine anti-EGFR monoclonal antibody cetuximab. Despite clear clinical importance, intrinsic or acquired resistance to EGFR inhibition is the rule rather than the exception. Currently, there is no predictive molecular marker for resistance or sensitivity to anti-EGFR therapy in HNSCC, including EGFR gene copy number as assessed in the EXTREME study. Given the poor prognosis and desperate lack of therapeutic options for patients with recurrent and/or metastatic HNSCC after failure of cetuximab, there is heightened interest in understanding resistance mechanisms in order to drive novel therapies for this population.

## 1.3 HGF/c-Met in Head and Neck Squamous Cell Carcinoma

An established intrinsic or acquired resistance mechanism to anti-EGFR therapy in HNSCC is primary or compensatory activation of alternate RTKs including c-Met. The *MET* oncogene encodes c-Met, an RTK bound exclusively by the ligand, hepatocyte growth factor (HGF). HGF is also known as "scatter factor;" this designation arose from early observations that HGF stimulates cellular decoupling and motogenesis. Overexpression of c-Met is transformative for normal cells and enhances motility, invasion/metastasis and angiogenesis. \*\* *MET* is an established driver of epithelial-to-mesenchymal transition, a phenotype associated with cetuximab resistance in HNSCC. \*\*16, 17

c-Met and/or HGF are overexpressed in ~80% of HNSCC,<sup>18</sup> and *MET* amplification has been reported in 13% of HNSCC tumors.<sup>19</sup> Moreover, several mutations have been identified in the *MET* oncogene in HNSCC, including alterations in the semaphorin ligand-binding, juxtamembrane, and RTK domains.<sup>19</sup> An activating point mutation (Y1253D) was described in 14% of patients in a Swiss chemoradiotherapy trial for locally advanced disease and predicted decreased metastasis-free survival, although the presence of this mutation in HNSCC was not confirmed in two whole-exome sequencing projects.<sup>20-22</sup>

Although validation and functional characterization of *MET* mutations in HNSCC is ongoing, the presence of *MET* overexpression, amplification, and mutation events suggests strong biologic relevance of this pathway. Furthermore, the current feasibility of measuring these events holds the promise that the clinical development of c-Met targeting in HNSCC may be accompanied by rational development of a predictive biomarker.

Of unique interest to the proposed study, the HGF/c-Met signaling pathway converges with the EGFR network at both the PI3K/Akt and MAPK nodes, suggesting the ability for reciprocal compensation. Several lines of evidence developed in our laboratories indicate that c-Met has an important role in resistance to EGFR based therapies. *In vitro*, the EGFR ligand TGF- $\alpha$  stimulated activation of c-Met in HNSCC cell lines, through prolonged tyrosine phosphorylation

and increased c-Met protein expression. Moreover, dual inhibition of EGFR (gefitinib) and c-Met (crizotinib) maximally inhibited phosphorylation of MAPK and Akt compared to single inhibition of either RTK, effectively abrogating crosstalk. Similarly, dual inhibition significantly reduced cell proliferation, invasion and wound healing, compared to mono- inhibition of either RTK. *In vivo*, dual inhibition of EGFR and c-Met retarded tumor growth, decreased the proliferative index, and enhanced apoptosis compared to either single agent.<sup>23</sup> A second laboratory found that dual blockade of c-Met (SU11274) and EGFR (erlotinib) in erlotinib-sensitive HNSCC cell lines decreased viability significantly more than exposure to either single agent, and isobologram indicated synergism.<sup>19</sup> Finally, growth factors have recognized potential to drive resistance to anticancer kinase inhibitors; in kinase addicted cell line models, the HGF ligand had broad potential to rescue kinase-addicted cancer cells dependent upon HER2 amplification, NRG1 autocrine stimulation, EGFR mutation, and BRAF mutation.<sup>24</sup> Finally, serum levels of HGF have been associated with resistance to EGFR inhibitors in *KRAS* wild-type metastatic colorectal cancer <sup>25</sup> and lung cancer <sup>25-27</sup>.

Above, convergent data suggest that HGF/c-Met pathway inhibition may overcome resistance to anti-EGFR therapy in R/M HNSCC, such as in patients with clinical cetuximab resistance. In theory, targeting HGF/cMet may have independent activity when administered as monotherapy in this setting, although this hypothesis has not been clinically tested. However, the cross talk and mutual compensation between c-Met and EGFR suggest that optimal benefit may be achieved by continuing cetuximab concurrent with HGF/c-Met pathway inhibition, in spite of established clinical resistance.

Ficlatuzumab (AV-299) is a humanized HGF-inhibitory immunoglobulin G1 (IgG1) monoclonal antibody that exhibits anti-tumor effects *in vitro* and in animal tumor models by 1) binding and neutralization of free HGF, 2) inhibition of c-Met phosphorylation, 3) inhibition of proliferation, 4) induction of apoptosis, and 5) inhibition of invasion and motility. Ficlatuzumab in combination with cetuximab resulted in prolonged tumor stasis/regression in 3 HNSCC xenograft models tested with increased activity compared to cetuximab alone in two of the three models tested. The recommended phase II dose (RP2D) for ficlatuzumab monotherapy has been established as 20 mg/kg IV every 2 weeks.

# 1.4 Phase Ib Study of the Combination of Ficlatuzumab and Cetuximab

We recently completed a phase Ib study of the combination of ficlatuzumab and cetuximab in patients with cetuximab-resistant, recurrent and/or metastatic HNSCC (NCT 02277197; Bauman JE et al, ASCO 2017). In this Narayana k-in-a-row phase I design, fixed-dose cetuximab was administered at 500 mg/m<sup>2</sup> IV every 2 weeks. Ficlatuzumab dose tiers were 10 mg/kg (starting

dose) or 20 mg/kg IV every 2 weeks (tier 2), with inter-patient escalation or de-escalation based on cumulative dose-limiting toxicities (DLT). The RP2D was set at dose tier 2 if no DLTs were observed after 8 enrolled patients, with expansion planned to n=12. Key eligibility criteria included: R/M HNSCC, cetuximab resistance (recurrence within 6 months of cetuximab-radiation or progression during/within 6 months of palliative cetuximab); ECOG performance status 0-1; mandatory baseline research biopsy. Candidate biomarkers included serum VeriStrat classification and tumor expression of pMet and HGF/cMet dimers.

From Sept 2015-June 2016, 12 pts were enrolled and treated. Primary site: 1 oral cavity; 3 oropharynx (1 p16+); 2 hypopharynx; 5 larynx; 1 external auditory canal. Platinum-refractory: 11/12. VeriStrat: 8 poor; 4 good. Three were treated at tier 1 and 9 at tier 2. No DLTs were observed. Grade 3 adverse events included: edema (1), hypoalbuminemia (1), infection (2), and thromboembolic event (2). Median PFS and OS at RP2D were 6.0 mos (90% CI = 2 mos – not reached) and 8.2 mos (90% CI = 2.7 mos – not reached), respectively. Response rate was 17% (90% CI = 0-28%): 2/12 partial response (PR); 1/3 at 10 mg/kg; 1/9 at 20mg/kg. Clinical benefit rate (PR + stable disease) was 67%. VeriStrat was not associated with PFS.

### 1.5 Study Rationale

Above, convergent data suggest that HGF/c-Met pathway inhibition may overcome resistance to anti-EGFR therapy in recurrent and/or metastatic HNSCC. The promising clinical activity observed in patients with cetuximab-resistant, recurrent and/or metastatic HNSCC during phase Ib compels further study in the same poor prognosis population. In theory, targeting HGF/cMet may have independent activity when administered as monotherapy in this setting, although this hypothesis has not been clinically tested. We also hypothesize that the cross talk and mutual compensation between c-Met and EGFR may necessitate the continuation of cetuximab with HGF/c-Met pathway inhibition, to optimize benefit. Thus we proposed a randomized, phase II study evaluating the efficacy of ficlatuzumab, with or without cetuximab, in patients with cetuximab-resistant, recurrent and/or metastatic HNSCC.

# 1.6 Ficlatuzumab (AV-299)

#### 1.6.1 Introduction

Ficlatuzumab (AV-299) is a humanized HGF inhibitory immunoglobulin G1 (IgG1) monoclonal antibody that exhibits anti-tumor effects in vitro and in animal tumor models by 1) binding and neutralization of free HGF, 2) inhibition of c-Met phosphorylation, 3) inhibition of proliferation, 4) induction of apoptosis, and 5) inhibition of invasion and motility.

Hepatocyte growth factor is the soluble ligand for the c-Met tyrosine kinase receptor. Hepatocyte growth factor/c-Met pathway dysregulation by over-expression or genetic alteration

is frequently observed in many types of cancer. Ficlatuzumab exhibited potent in vivo inhibitory activity in autocrine and paracrine xenograft models as single agents in GBM, multiple myeloma and RCC. Ficlatuzumab demonstrated enhanced antitumor activity when combined with targeted therapy or chemotherapy, such as erlotinib, cetuximab, tivozanib or temozolomide in a panel of xenograft models, suggesting ficlatuzumab may have anti-tumor activity in multiple tumor indications. Ficlatuzumab in combination with cetuximab resulted in prolonged tumor stasis/regression in all 3 HNSCC xenograft models tested with increased activity compared to cetuximab alone in two of the three models tested

A summary of ficlatuzumab's pertinent efficacy results and safety data follow. Please refer to the ficlatuzumab Investigator Brochure (IB) for descriptions of all available data.

### 1.6.2 Ficlatuzumab clinical experience

An overview of the clinical data available for ficlatuzumab clinical studies; protocols P05538 (phase I), P05670 (pharmacodynamic study) and P06162 (phase Ib/II in NSCLC) is provided below. Final data for Protocols P05538 (with the exception of the 1 ongoing subject) and P05670 and preliminary data for Protocol P06162 are included in the Ficlatuzumab Investigator Brochure.

Protocol P05538 includes data for 41 subjects diagnosed with relapsed or refractory solid tumors that were metastatic or unresectable, or symptomatic relapsed or refractory multiple myeloma. There were 7 cohorts in total. The dose-escalation cohorts included subjects diagnosed with relapsed or refractory solid tumors that were metastatic or unresectable that were treated at the following dose levels: Cohort 1 (2 mg/kg), Cohort 2 (5 mg/kg), Cohort 3 (10 mg/kg), and Cohort 4 (20 mg/kg); safety expansion Cohort 5 (20 mg/kg, which was the RP2D). The additional cohorts were the Erlotinib Combination Cohort (ficlatuzumab 20 mg/kg and erlotinib 150 mg) and Multiple Myeloma Cohort (ficlatuzumab 20 mg/kg). There were 24 subjects enrolled in the dose escalation/safety expansion cohorts, 13 subjects enrolled in the Erlotinib Combination Cohort, and 4 subjects enrolled in the Multiple Myeloma Cohort. After an interim review of the data, there was no signal of clinical benefit to subjects with multiple myeloma; therefore, enrollment into this cohort was terminated.

Protocol P05670 was a pharmacodynamic study including data for 19 subjects with advanced solid tumors and liver metastases. There were 3 dose cohorts of ficlatuzumab (2, 10, and 20 mg/kg). Six subjects were enrolled in the Dose Level 1 Cohort (2 mg/kg), 7 subjects were enrolled in the Dose Level 2 Cohort (10 mg/kg), and 6 subjects were enrolled in the Dose Level 3 Cohort (20 mg/kg). The best responses in the study were stable disease seen 5/18 patients and the median duration of treatment was 6 weeks. The Pk of ficlatuzumab was characterized by low

clearance and a half-life of 7-10 days. Ficlatuzumab treatment at 20 mg/kg, but not at 2 and 10 mg/kg, demonstrated pharmacodynamic modulation in the tumor by inhibiting HGF/c-Met pathway and downstream signaling for cell proliferation, survival, and angiogenesis in majority of the patients treated.

Protocol P06162 is a Phase 1b/2 study including preliminary data for 199 subjects. Phase 1b enrolled Asian subjects with NSCLC or other advanced solid tumors. Phase 2 enrolled Asian subjects (nonsmokers or light ex-smokers) with previously untreated lung adenocarcinoma. Subjects in Phase 1b are treated with a dose of ficlatuzumab 10 mg/kg or 20 mg/kg in combination with gefitinib 250 mg. Subjects in Phase 2 are treated with a combination of ficlatuzumab 20 mg/kg and gefitinib 250 mg or gefitinib 250 mg monotherapy. Upon progression in the gefitinib monotherapy arm, subjects who initially demonstrated disease control with single agent gefitinib were offered to receive the combination of ficlatuzumab 20 mg/kg and gefitinib 250 mg, provided that safety was maintained and the subject continued to meet eligibility criteria. There were 15 subjects enrolled in Phase 1b (3 subjects enrolled in the 10 mg/kg cohort and 12 subjects enrolled in the 20 mg/kg) and 184 subjects enrolled in Phase 2 (90 subjects enrolled in the Combination Cohort and 94 subjects enrolled in the Gefitinib Monotherapy Cohort). Of the subjects enrolled in the Phase 2 Gefitinib Monotherapy Cohort, 20 were crossed over to receive the combination of ficlatuzumab 20 mg/kg and gefitinib 250 mg.

The addition of ficlatuzumab to gefitinib did not result in a significant improvement in ORR (primary endpoint) or PFS in the intent to treat population. The ficlatuzumab/gefitinib combination demonstrated a trend for increased ORR and OS in a subset of patients without EGFR sensitizing mutations and increased PFS, OS and ORR in a subset of patients with high stromal HGF. Overall survival data continues to mature and are being analyzed in the intent to treat group as well as other biomarker subsets. The combination of ficlatuzumab and gefitinib was well tolerated in this patient population.

## 1.6.3 Ficlatuzumab Safety Experience

Refer to the Aveo Pharmaceuticals Investigator Brochure for the most up-to-date information.

Data from the first-in-human dose-escalation study (Study P05538) in 41 subjects diagnosed with relapsed or refractory solid tumors or lymphoma that was metastatic or unresectable, or symptomatic relapsed or refractory multiple myeloma showed ficialtuzumab to be well-tolerated as monotherapy at the 4 dose levels tested (2, 5, 10 or 20 mg/kg) and in combination with erlotinib (20 mg/kg ficialtuzumab and 150 mg/day erlotinib). The maximum administered dose of 20 mg/kg intravenous (IV) ficialtuzumab every 2 weeks as monotherapy and in combination with erlotinib (150 mg/day) was determined to be the RP2D.

There were no DLTs observed with single-agent ficlatuzumab. One subject in the ficlatuzumab plus erlotinib combination cohort experienced a Grade 3 mucositis which the investigator determined was possibly related to ficlatuzumab and related to erlotinib. The most common treatment-emergent adverse events (TEAEs) were fatigue (18 subjects, 44%), peripheral edema (13 subjects, 32%), hypokalemia (11 subjects, 27%), and nausea (10 subjects, 24%). The most frequently reported related TEAEs were fatigue (12 subjects [29%]; 9 subjects monotherapy [22%], 3 subjects erlotinib combination [7%]); peripheral edema (6 subjects [15%]; 5 subjects monotherapy [12%], 1 subjects erlotinib combination [2%])); headache (5 subjects [12%]; 4 subjects monotherapy [10%], 1 subjects erlotinib combination [2%]), pruritus (5 subjects [12%]; 3 subjects monotherapy [7%], 2 subjects erlotinib combination [5%]), and rash maculo-papular (5 subjects [12%]; 5 subjects erlotinib combination [12%]).

Serious adverse events (SAEs) considered at least possibly related to ficlatuzumab included Grade 1 blindness transient, Grade 4 hyperkalemia, and Grade 1 hypokalemia, one case each.

Data from a Phase 1 pharmacodynamic study (Study P05670) in 19 subjects with advanced solid tumors and liver metastases showed ficlatuzumab to be well-tolerated as monotherapy at the 2 to 20 mg/kg dose range tested. There were no DLTs in this study. The most frequently reported TEAEs were asthenia, peripheral edema, and hepatic pain (each reported by 6 subjects [32%]), and cough (5 subjects [26%]). The only related adverse event (AE) was pyrexia, which occurred in 1 subject in the 2 mg/kg treatment group (5%). There were no SAEs considered at least possibly related to ficlatuzumab.

The safety profile of ficlatuzumab was acceptable and similar to the drugs in its class. Serum albumin decreased to below the lower limit of normal at end of study for all exposed subjects. Serum albumin levels began to recover at the follow up visit.

Data from the Phase 1b portion of the Study P06162 in 15 subjects with non-small cell lung cancer (NSCLC) showed ficiatuzumab to be well-tolerated in combination with gefitinib. Ficiatuzumab at 20 mg/kg plus gefitinib at 250 mg/day was determined to be the RP2D.

Of the 12 Phase 1b subjects who received the RP2D, 2 subjects (17%) had DLTs: an SAE of diffuse alveolar damage in 1 subject that resulted in death, and Grade 3 acneiform dermatitis in 1 subject. Both of these events were assessed by the investigator as probably related to gefitinib and/or ficialtuzumab.

The most common TEAEs were dermatitis acneiform (in 10 subjects [67%]), decreased appetite (7 subjects [47%]), diarrhea (6 subjects [40%]), and cough, fatigue, and paronychia (each in 5

subjects [33%]). The most frequently reported study drug-related TEAEs were dermatitis acneiform (10 subjects [67%]), paronychia (5 subjects [33%]), and diarrhea (4 subjects [27%]).

Ficlatuzumab monotherapy has been generally well tolerated. <u>Table 1</u> lists the TEAEs that, based upon preliminary monotherapy safety data, could be reasonably assumed to be associated with ficlatuzumab.

Data from the Phase 2 portion of the Study P06162 in 184 subjects with non-small cell lung cancer (NSCLC) showed ficiatuzumab to be well tolerated in combination with gefitinib. <u>Table 2</u> lists the preliminary data on TEAEs with  $a \ge 10\%$  difference between the two treatment groups (ficiatuzumab+gefitinib vs gefitinib monotherapy).

**Table 1: Adverse Events Expected to Occur with Ficlatuzumab Monotherapy** 

| MedDRA Preferred Term |
|---|
| Decreased appetite |
| Diarrhea |
| Dry skin |
| Edema peripheral |
| Fatigue |
| Headache |
| Hypoalbuminemia |
| Hypokalemia |
| Hypomagnesemia |
| Myalgia |
| Nausea |
| Pruritus |
| Rash |
| Chills |
| Dizziness |
| Muscle Spasms |
| Bacterial skin infection, which may cause swelling, redness, and sensitivity |
| Vomiting |

MedDRA = Medical Dictionary for Regulatory Activities

**Table 2: TEAEs w/ ≥ 10% Difference between Treatment Groups (Study P06162)** 

| TEAE, n (%) | Ficlatuzumab<br>n=9 | | Gefitinil<br>n=9 | |
|---|---|---|---|---|
| | All grades | Grade 3 | All grades | Grade 3 |
| Paronychia | 42 (47) | - | 23 (25) | 1 (1) |
| Acne | 24 (27) | 1 (1) | 15 (16) | - |
| Peripheral edema | 34 (38) | 2 (2) | 4 (4) | 1 (1) |
| Dizziness | 17 (19) | - | 8 (9) | - |
| Eczema | 15 (17) | 2 (2) | 7 (7) | - |
| Hypoalbuminemia | 18 (20) | 2 (2) | 3 (3) | - |
| Gingival bleeding | 11 (12) | - | 1 (1) | - |

Ficlatuzumab has not been found to be immunogenic in any patients treated to date; no post-treatment anti-drug antibodies have developed.

#### 1.7 Cetuximab

#### 1.7.1 FDA Indications in HNSCC

Cetuximab is an IgG1, chimeric murine-human antibody against EGFR that was first approved by the U.S. Food and Drug Administration for the treatment of patients with recurrent and/or metastatic HNSCC in 2006. As cetuximab is a common and accepted standard of care, commercial cetuximab will be used in this study. Please see the cetuximab package insert for complete prescribing information (<a href="http://pi.lilly.com/us/erbitux-uspi.pdf">http://pi.lilly.com/us/erbitux-uspi.pdf</a>).

The most common adverse events (≥25%) associated with cetuximab in clinical trials include: cutaneous adverse reactions (acneiform rash, pruritus, and nail changes), headache, diarrhea, hypomagnesemia/accompanying electrolyte abnormalities, and infection.

The most serious adverse reactions associated with cetuximab are: infusion reactions, cardiopulmonary arrest, dermatologic toxicity and radiation dermatitis, sepsis, renal failure, interstitial lung disease, and pulmonary embolus.

#### 1.7.2 Rationale for Every Two Week Dosing Schedule of Cetuximab

The early studies that established weekly dosing of cetuximab did not establish an MTD.<sup>28, 29</sup> Subsequent pharmacokinetic studies were conducted in patients with advanced colorectal cancer, exploring other doses and schedules. In studies of q2week dosing, cetuximab doses of 400 to 700 mg/m2 q2weeks were well tolerated and the MTD was not reached.<sup>30</sup> Pharmacokinetic analysis showed that trough cetuximab levels for the 500 mg/m² q2weeks, 600 mg/m² q2weeks, and 250 mg/m² weekly regimens were comparable.<sup>30, 31</sup> Pharmacodynamic

studies, in which subjects underwent skin biopsies at baseline and at week 4 showed that all cetuximab dose levels yielded comparable changes in the expression of pEGFR, pMAPK, Ki67, p27, and pSTAT3 as detected with immunohistochemistry.<sup>32</sup> Cetuximab at 500 mg/m<sup>2</sup> q2weeks was identified as a convenient and feasible dose.

In recurrent and/or metastatic HNSCC, a randomized phase II study compared two q2week cetuximab doses and found that the dose of 500 mg/m²/q2weeks resulted in similar efficacy to weekly dosing at 250 mg/m²/week, with no therapeutic advantage for 750 mg/m² q2weeks. Due to convenience and comparable efficacy, clinical trials in HNSCC are now integrating the q2week dosing schedule.<sup>33</sup>

## 1.8 Correlative Studies Background

# 1.8.1 Tumoral Activation of HGF/cMet Pathway

We have published a report of a cohort of 56 HNSCC patients with tumor protein levels of HGF and cMet calculated by the H score (intensity weighted by percent tumor).<sup>18</sup> We found that HNSCC tumors overexpress both HGF and c-Met as compared to adjacent tissue, as demonstrated below in Figure 1. Ongoing work indicates a bidirectional positive feedback loop between tumor-associated fibroblasts (TAF) which secrete HGF, and HNSCC tumor cells whose conditioned media stimulate HGF secretion from TAFs.<sup>34</sup> In a preclinical HNSCC-TAF co-culture model, ficlatuzumab inhibited HNSCC progression via reduced cMet and mitogen-activated protein kinase (MAPK) signaling.<sup>35</sup>

During the phase Ib trial evaluating the combination of ficlatuzumab and cetuximab in patients with cetuximab-resistant, recurrent and/or metastatic HNSCC, we evaluated three candidate baseline biomarkers for feasibility and relationship to response: VeriStrat; tumoral expression of pMet; and tumoral expression of HGF/cMet dimers. There was no relationship between VeriStrat status and PFS. pMet and HGF/cMet dimer analyses are pending.



**Figure 1:** HGF and c-Met are overexpressed in head and neck cancer. HGF and c-Met protein levels were assessed by immunohistochemistry in HNSCC tumors and paired adjacent mucosa (n = 26). Intensity (integer scale 0 to +3) and percent of tumor stained were evaluated. A weighted score of intensity times percent of tumor stained was calculated. A, tumor tissues showed increased HGF and c-Met staining compared with paired adjacent mucosal tissues. B, two-tailed Wilcoxon signed-rank test for paired samples indicated significant differences in weighted HGF and c-Met intensity in tumor versus paired adjacent mucosa (HGF; P < 0.001; c-Met; P = 0.04). C, HGF and c-Met immunohistochemistry score frequency distributions indicate that higher levels of HGF are more frequently present in HNSCC tumors than c-Met.<sup>18</sup>

In this clinical trial, patients will undergo a research biopsy at baseline. We will investigate the relationship between candidate biomarkers and clinical outcomes on each arm, including the following:

- Dimers (Monogram assay): HGF/cMet, EGFR/EGFR, EGFR/HER2
- Signaling proteins: pMet, bFGF, pMAPK, pAkt

We will also analyze HGF and cMet in archived diagnostic biopsies which took place before clinical cetuximab exposure, as available.

# 1.8.2 Peripheral Biomarkers of HGF/cMet Pathway Activation

We will also assess candidate peripheral biomarkers for relationship to clinical outcomes. In the present study, we will evaluate candidate peripheral biomarkers related to HGF/c-Met pathway

activation, including:

- HGF
- Soluble HGF
- IL6

### 1.8.3 Genomic Alterations: PIK3CA, PTEN, and HRAS

The mutational landscape of HNSCC was assessed by whole exome sequencing of 74 tumor-normal pairs.<sup>37</sup> Several mutations in HNSCC interact with the EGFR and HGF/c-Met signaling pathways and may modulate the impact of pathway antagonism. These include *PIK3CA* (8%), *PTEN* (8%), and *HRAS* (4%) mutations. As we did not confirm the presence of activating *MET* mutations or amplification described by others, and the TCGA has demonstrated less than 1% prevalence in >300 case of *MET* mutation or *MET* amplification, we will not assess *MET* mutation or amplification status.<sup>19</sup>.<sup>38</sup>

#### 1.8.4 Immune Biomarkers

HNSCC is an immunosuppressive disease. Patients demonstrate lower absolute lymphocyte counts than healthy subjects <sup>39</sup>, impaired natural killer (NK) cell activity <sup>40, 41</sup>, and poor antigen-presenting function <sup>42, 43</sup>. Mechanistically, HGF inhibits dendritic cell activation by blocking IκB kinase activity and subsequent nuclear factor-κB activation. Inhibition of IκB kinase is mediated by HGF-induced activation of c-Src.<sup>44</sup> Bruton's tyrosine kinase is also necessary for the association of c-Src with c-Met.<sup>45</sup>

We will evaluate and describe the immune infiltrate in both archived biopsies (prior to cetuximab exposure) and the baseline research biopsies (after cetuximab resistance) from patients enrolled in this study. We will relate immunoscores to clinical outcomes.

## 1.8.5 Patient-Reported Outcomes

Quality of Life (QOL). The Functional Assessment of Cancer Therapy-Head and Neck Symptom Index (FACT-H&N SI) will be used to measure global quality of life and functional decline from the patient's perspective. The FACT-H&N SI is an internationally validated QOL tool. It is a multidimensional, patient-self report QOL instrument that has been specifically designed and validated for this patient population.<sup>46</sup> The questionnaire consists of 10 core items that assess patient function in 4 domains: Physical, Social/Family, Emotional, and Functional well-being. Each item is rated on a 0 to 4 Likert type scale, and then combined to produce subscale scores for each domain, as well as a global QOL score; higher scores represent better QOL. The FACT-H&N SI can be completed by the patient in about 5 minutes, is available in 26 languages, and will be completed at baseline, end of cycle 2, and end of cycle 6. See Appendix A for FACT-H&N-SI.

# 2. STUDY OBJECTIVES

## 2.1 Primary

To assess the efficacy of ficlatuzumab, with or without concurrent cetuximab, in patients with cetuximab-resistant, recurrent and/or metastatic HNSCC as measured by Progression-Free Survival (PFS).

### 2.2 Secondary

- To describe toxicity
- To evaluate response rate and overall survival in both treatment arms.

## 2.3 Exploratory

- To describe patient-reported quality of life.
- To evaluate the relationship between clinical outcomes (Progression-Free Survival and Response Rate) and candidate tumoral, genomic, peripheral, and immune biomarkers, potentially including but not limited to:
  - Tumor HGF and cMet expression
  - mutations in PIK3CA, PTEN, and HRAS;
  - o peripheral serum biomarkers including HGF, soluble HGF, and IL6;
  - peripheral lymphocyte populations;
  - o archived and baseline immune infiltrate;
  - tumor HPV status.

#### 3. PATIENT SELECTION

#### 3.1 Inclusion Criteria

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

- Patients must have histologically confirmed HNSCC from any primary site, except nasopharyngeal if WHO Type III (non-keratinizing and EBV-positive).
  - Eligible histologies include:
    - Basaloid, poorly differentiated, and undifferentiated carcinoma histologies.
    - Nasopharyngeal carcinoma, WHO Type I and II (keratinizing, non-EBV positive).
    - Paranasal sinus, lip, and external auditory canal sites.

 Squamous cell carcinoma of unknown primary, clearly related to the head and neck.

**Note:** Documentation of primary site diagnosis must be submitted with the registration request.

- Patients must have recurrent and/or metastatic disease, fulfilling at least one of the criteria defined below:
  - Incurable disease as assessed by surgical or radiation oncology;
  - Metastatic (M1) disease;
  - Persistent or progressive disease following curative-intent radiation, and not a candidate for surgical salvage due to incurability or morbidity. **Note:** Patients who decline radical surgery are eligible.
- For patients with **oropharyngeal primary site** or **unknown primary site** only: Patients must have known tumoral HPV status (p16). (Acceptable standards include p16 immunohistochemistry (where a tumor is classified as p16-positive when showing diffuse nuclear and cytoplasmic staining in at least 70% of tumor cells) and/or assessment of HPV DNA.)

**Note:** For these subjects, documentation of p16 status must be submitted with the registration packet.

- Patients must be cetuximab-resistant by fulfilling at least one of the two criteria defined below:
  - Disease persistence or recurrence within 6 months of completing definitive radiotherapy with concurrent cetuximab for locally advanced disease. Induction chemotherapy, if given, may or may not have included cetuximab.
  - Disease progression during, or within 6 months, of cetuximab treatment in the recurrent and/or metastatic setting.

**Note:** Prior cetuximab exposure may have occurred in any line of therapy (first line, second line, etc.) and is not required to be the most recent therapy received.

- Patients must be platinum-resistant or platinum-ineligible by fulfilling at least one of the three criteria defined below:
  - Disease persistence or recurrence within 6 months of completing definitive radiotherapy for locally advanced disease, where platinum chemotherapy was administered as a component of induction and/or concurrent systemic treatment.
  - Disease progression during, or within 6 months, of treatment with platinum chemotherapy (e.g., carboplatin or cisplatin) in the recurrent and/or metastatic setting.

 The patient is not an acceptable candidate for platinum chemotherapy due to medical comorbidities, in the judgment of the local investigator.

**Note:** Prior platinum exposure may have occurred in any line of therapy (first line, second line, etc.) and is not required to be the most recent therapy received.

 Patients must have prior exposure to an anti-PD1 or anti-PDL1 mAb, if eligible for immunotherapy in the judgment of the local investigator.

**Note:** Prior exposure to investigational immunotherapies, including anti-CTLA4, anti-OX40, anti-CD40, anti-CD27, anti-TNFR antibodies or other investigational immunotherapies, is acceptable.

- Patients must have Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 at time of informed consent (see Appendix B).
- Patients must be age ≥ 18 years.
- Patients must consent to a research biopsy of tumor tissue at baseline, for conduct of
  correlative studies. In cases where a fresh biopsy is not feasible (i.e., if an accessible
  tumor site cannot be biopsied with acceptable clinical risk), archival tissue may be
  submitted instead, after discussion with and approval by the Sponsor-Investigator.
- Patients must have measurable disease per RECIST criteria, version 1.1 (see <u>Section 6</u>) per scan within 28 days prior to registration.
- Patients must have adequate electrolytes, liver, renal, and hematology function as defined below within 28 days of registration:
  - o Absolute neutrophil count (ANC) ≥ 1500/mm<sup>3</sup>
  - Platelet count (PLT)  $\geq$  75,000/mm<sup>3</sup>
  - o Creatinine clearance ≥ 30 mL/min per estimated by the Cockraft-Gault formula:
    - Calculated Creatinine Clearance = [(140-age) X (actual body weight in kg) X (0.85 if female)]/(72 X serum creatinine)
  - o Total bilirubin ≤ 1.5 times upper-limit of normal (ULN)
  - AST (aspartate aminotransferase) ≤ 3 times ULN
  - ALT (alanine aminotransferase) ≤ 3 times ULN
  - Magnesium ≥ 1.2 mg/dL or 0.5 mmol/L\*
  - Corrected Calcium ≥ 8.0 mg/dL or 2.0 mmol/L\*
  - Potassium ≥ 3.0 mmol/L\*
  - Serum albumin  $\geq$  25 g/L ( $\geq$  2.5 g/dL)

(\***Note:** Patients may be supplemented to achieve acceptable electrolyte values.)

- Patients must sign written informed consent prior to beginning study screening procedures. Patients must have the ability to understand and the willingness to sign a written informed consent document.
- Women of child-bearing potential (WOCBP) must agree to have a pregnancy test within 14 days prior to registration and a repeated test within 3 days of the first dose of ficlatuzumab.
- Patients must agree to use highly effective contraceptive measures while on study and for 60 days after the last dose of study drug. This includes: Men of reproductive potential AND women of childbearing potential.
  - o Effective birth control includes (a) intrauterine device (IUD) plus one barrier method; or (b) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm).

#### 3.2 Exclusion Criteria

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

- Nasopharyngeal primary site if WHO Type III (non-keratinizing and EBV-positive as established at the local site).
- History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational agent.
- Prior treatment with an HGF/cMet inhibitor such as rilotumumab, crizotinib, MetMAb, or ARQ197.
- Uncontrolled central nervous system (CNS) metastases, including leptomeningeal metastases, are not allowed.

**Note:** Subjects with previously treated brain metastases will be allowed if the brain metastases have been stable without steroid treatment for at least 2 weeks (radiotherapy or surgery).

- Failure to recover to Grade 1 or baseline from all toxic effects of previous chemotherapy, radiation therapy, biologic therapy, immunotherapy, and/or experimental therapy, with the exception of:
  - Alopecia,
  - Grade ≤ 2 peripheral neuropathy,
  - Grade ≤ 2 cetuximab-related rash or other skin changes,
  - o Hypomagnesemia (acceptable values detailed in the exclusion criteria below),
  - o Hypokalemia (acceptable values detailed in the exclusion criteria below), and

- The acceptable ANC and PLT inclusion criteria values above.
- Treatment with cetuximab 2 weeks prior to the first dose of study drug. A washout period of 2 weeks from prior cetuximab is required if applicable.
- Treatment with cytotoxic chemotherapy, targeted therapy, immunotherapy or investigational drug 3 weeks prior to the first dose of study drug. A washout period of 3 weeks from any prior cytotoxic chemotherapy, targeted therapy, immunotherapy or investigational drug is required, if applicable.
- Significant underlying pulmonary disease, including pulmonary hypertension or interstitial pneumonitis.
- Peripheral edema ≥ Grade 2 per NCI-CTCAE version 4.0.
- Significant cardiovascular disease, including:
  - o Cardiac failure New York Heart Association (NYHA) class III or IV.
  - Myocardial infarction within 6 months prior to registration.
  - Severe or unstable angina within 6 months prior to registration.
  - History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation).
  - Cardiac arrhythmia requiring anti-arrhythmic medication(s). (Beta-blockers, calcium channel blockers, and digoxin administered for the purpose of rate control of supraventricular tachycardia, including atrial fibrillation and atrial flutter, are not classified as anti-arrhythmic medications for purposes of trial eligibility.)
- Significant thrombotic or embolic events within 28 days prior to registration. (Significant thrombotic or embolic events include but are not limited to stroke or transient ischemic attack (TIA). Catheter-related thrombosis is not a cause for exclusion. Diagnosis of deep vein thrombosis or pulmonary embolism is allowed if it occurred > 28 days prior to registration and the patient is asymptomatic and stable on anti-coagulation therapy.)
- Any other medical condition (e.g., alcohol abuse) or psychiatric condition that, in the opinion of the local Investigator, might interfere with the subject's participation in the trial or interfere with the interpretation of trial results.
- History of second malignancy within 2 years prior to registration except:
  - o Excised and cured non-melanoma skin cancer,
  - Carcinoma in situ of breast or cervix,
  - Superficial bladder cancer,
  - Stage I differentiated thyroid cancer that is resected or observed,
  - pT1a /pT1b prostate cancer comprising < 5% of resected tissue with normal prostate specific antigen (PSA) since resection, or

- cT1a/cT1b prostate cancer treated with brachytherapy or external beam radiation therapy with normal PSA since radiation.
- Not completely recovered from any previous surgery.

**Note:** Complete recovery is in the opinion of the treating investigator. Consult the Sponsor-Investigator, if needed.

Active systemic infection requiring systemic antibiotics or antifungals within 7 days prior
to first dose of study drug, except tetracycline family antibiotics (tetracycline,
doxycycline, minocycline) administered for the management of cetuximab-related rash
may be continued per the Investigator's judgment.

**Note:** Active topical infections (for example oral thrush) do not exclude a subject even if treated with systemic antibiotics or systemic antifungals.

- History of severe infusion reaction to cetuximab or a monoclonal antibody.
- Known to be HIV positive. Note: HIV testing is not required for entry into this protocol.
- Women who are pregnant or breastfeeding. (A negative urine pregnancy test must be confirmed within 14 days of registration and repeated within 3 days of the first dose of study drug.)

#### 4. PATIENT REGISTRATION AND RANDOMIZATION

#### 4.1 Registration

After eligibility has been confirmed, registration will be submitted to the University of Arizona Cancer Center using the Registration Form. The study Eligibility Checklist and Registration Form, with required source documentation must be provided for the randomization. The following source documentation must be submitted and other documentation may be requested:

- Confirmation of primary site diagnosis.
- For oropharyngeal primary site or unknown primary site, confirmation of p16 (HPV) status.
- Signed consent page with Subject ID added, and PHI redacted.

#### 4.2 Randomization

Subjects will be randomized to one of the following two arms:

- Arm A: Ficlatuzumab monotherapy, or
- Arm B: Ficlatuzumab + cetuximab combination therapy.

Randomization will be performed by the UACC Biostatistics Shared Resource.

#### Stratification Factors:

Patients will be stratified by HPV status, a known prognostic factor in recurrent and/or metastatic HNSCC, and study center.

- HPV-positive vs. HPV-negative as assessed by p16 status.
  - To be classified as HPV-positive, patients must meet BOTH of the following criteria:
    - 1) either oropharynx or unknown primary site; AND
    - 2) p16+ by immunohistochemistry, where ≥ 70% of tumor cells demonstrate diffuse nuclear and cytoplasmic staining with p16 antibody.
  - For purposes of stratification, the remainder of patients will be classified as HPVnegative.
- Study Center

#### 5. TREATMENT PLAN

Note: One cycle consists of 28 days (with a window of +7 days, that is 35 days maximum), and includes two doses of study drug(s), on Day 1 and Day 15 (+/- 3 days unless there is a delay as described in <u>Section 5.5</u>).

The doses of both ficlatuzumab and cetuximab will be recalculated **only if** there is a  $\geq$  10% change in weight. Exception: If, in the opinion of the treating investigator, weight change of  $\geq$  10% is due to edema, recalculation of the ficlatuzumab dose is not required. This decision must be clearly documented.

Refer to <u>Section 5.5</u> for additional information on dose modifications, delays and skipped treatments, and treatment stoppage rules.

Treatment holidays are allowed, per investigator judgement. For the purposes of the study schedule, treatment holidays will be considered skipped doses.

#### 5.1 Ficlatuzumab

The ficial fiction and administration information.

The lot of ficlatuzumab will expire on March 31, 2021. The latest administration of ficlatuzumab will be on or before that date. Subjects on the treatment portion of the trial at that time will stop the study treatment and be censored for progression. Subjects will be followed for AEs per

<u>Section 8.5.1</u>, then enter the progressive disease follow-up as described in <u>Section 5.4.1</u> and <u>Section 8.5.3</u>. Investigators will discuss the transition with their subjects in a timely manner prior to the expiration.

#### **5.1.1** Route of Administration

Ficlatuzumab will be administered as an IV infusion.

#### 5.1.2 Dose and Schedule

Ficlatuzumab will be administered at the dose of 20 mg/kg IV every 2 weeks (+/- 3 days). Ficlatuzumab will be administered over 30-60 minutes.

Ficialty amab dose must be recalculated if there is a  $\geq$  10% change in weight. Exception: If, in the opinion of the treating investigator, weight change of  $\geq$  10% is due to edema, recalculation of the ficialty amab dose is not required. This decision must be clearly documented.

Protocol-specified dose modifications are permitted. See <u>Table 3</u> below for dose reduction levels.

#### **5.1.3 Order of Administration for Arm B (Combination Arm)**

Subjects randomized to the combination arm will receive cetuximab and ficial fiction on the same day. Cetuximab will be administered first per the dose and schedule described in <u>Section 5.2.2</u>. Ficial will be administered 30-60 minutes after the completion of the cetuximab infusion, per the dose and schedule described in <u>Section 5.1.2</u>.

#### 5.2 Cetuximab

#### 5.2.1 Route of Administration

Cetuximab will be administered as an IV infusion.

#### 5.2.2 Dose and Schedule

Cetuximab will be administered at the dose of 500 mg/m<sup>2</sup> IV every 2 weeks (+/- 3 days), on the same day as ficlatuzumab. Suggested schedule:

- The first dose will be administered over 120 minutes (+/- 15 minutes) and at a rate no faster than 10 mg/minute.
- Subsequent doses will be infused at a rate no faster than 10 mg/minute.

Local standard of care can be followed if it is different than this suggested schedule.

Cetuximab dose must be recalculated if there is a  $\geq$  10% change in weight. Exception: If, in the opinion of the treating investigator, weight change of  $\geq$  10% is due to edema, recalculation of the ficlatuzumab dose is not required. This decision must be clearly documented.

Protocol-specified dose modifications are permitted. See <u>Table 3</u> below for dose reduction

levels.

## 5.2.3 Order of Administration for Arm B (Combination Arm)

See Section 5.1.3.

#### 5.2.4 Premedications

Prior to the first dose of cetuximab, 50 mg of diphenhydramine will be administered PO or IV. If the patient shows no evidence of hypersensitivity, the dose of diphenhydramine may be reduced to 25 mg PO or IV, or eliminated, per investigator judgment. In patients intolerant of diphenhydramine, a non-sedating antihistamine (eg. cetirizine 10 mg) may be substituted per local preference. Alternately or in addition, a dose of IV steroids (eg. dexamethasone 10 mg; hydrocortisone 50 mg) may be substituted per local preference.

## **5.3 General Concomitant Medication and Supportive Care Guidelines**

<u>Colony-Stimulating Factors</u>: Colony stimulating factors, including G-CSF, pegylated G-CSF, and erythropoietin analogs may be used in accordance with local and national practice guidelines.

## 5.4 Duration of Treatment and Follow-up

### 5.4.1 Treatment Duration:

Treatment will continue until one of the following criteria applies:

- Disease progression,
- Intercurrent illness that prevents further administration of treatment,
- Unacceptable adverse event(s),
- Patient elects to withdraw from the study for any reason,
- General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator, including pregnancy.
- March 31, 2021 (expiration date of ficlatuzumab)

#### 5.4.2 Follow up duration - WITHOUT progressive disease:

Patients who stop treatment **without** progressive disease will be followed approximately every 8 weeks (+/- 2 weeks) until progression of disease, then every 12 weeks (+/- 2 weeks) for 2 years after disease progression. Patients who begin a new line of therapy will be censored for progression and be followed per the progressive disease schedule. Refer to <u>Section 8.5</u> for post-treatment protocol-required evaluations.

## 5.4.3 Follow up duration - WITH progressive disease:

Patients who stop treatment **with** progressive disease will be followed for survival every 12 weeks (+/- 2 weeks) for two years after disease progression, or until death, whichever occurs first. Refer to Section 8.5 for post-treatment protocol-required evaluations.

### 5.4.4 Follow up for unacceptable adverse events

Patients who stop the study treatment for unacceptable adverse event(s) will be followed for 60 days after the last dose of study drug or until resolution or stabilization of the unacceptable adverse event. Patients will then be followed per the schedule described in <u>Section 5.4.2</u> (also see <u>Section 8.5</u>).

### **5.5 Dose Delays and Modifications**

### 5.5.1 Treatment Plan Interruptions and Delays

Treatment delays and/or skipped visits must be implemented as follows.

These definitions are independent of the +/- 3-day window for treatment visits.

- Treatment delays: Treatment delayed 7 or less days will be considered a delay.
- Skipped/missed treatments: For a treatment delay that is more than 7 days, the treatment will be considered a missed/skipped visit and the next treatment should occur at the next regularly scheduled visit.

Note regarding multiple delays within 2 cycles: Two or more delays within 2 cycles may result in the every-8-week scan occurring out of window. Contact the Sponsor-Investigator team for consensus on subsequent scheduling.

#### 5.5.2 Dose Reduction Levels

The following table summarizes dose levels available for protocol-specified dose reductions of ficiatuzumab and/or cetuximab (Table 3).

**Table 3: Dose Reduction Levels** 

| Dose Level | Ficlatuzumab | Cetuximab |
|------------|------------------|-------------------------------|
| -1 | 15 mg/kg q2weeks | 400 mg/m <sup>2</sup> q2weeks |
| -2 | 10 mg/kg q2weeks | 300 mg/m² q2weeks |

Subjects may have up to two dose reductions. Subjects at the lowest ficial ficial dose level (10mg/kg) who experience an attributable Grade 3 or 4 toxicity will be discontinued from ficial ficial field benefit, a subject may resume treatment at 10 mg/kg after the AE has resolved or ameliorated to  $\leq$  Grade 2 or baseline. Contact the Sponsor-Investigator for consensus on subsequent treatment.

If a cetuximab-related toxicity results in discontinuation of cetuximab permanently, treatment with ficialty umab can continue.

If a ficlatuzumab-related toxicity results in discontinuation of ficlatuzumab permanently, per

discretion of the treating investigator, treatment with cetuximab can continue.

# **5.5.3 Treatment Stoppage Rules For Toxicity**

If any observed toxicity at least possibly related to ficlatuzumab and/or cetuximab prevents dosing within the scheduled study visit window, the dose for that study visit will be skipped and the next study drug administration will occur at the next scheduled dose. If a ficlatuzumab-related toxicity results in 2 consecutive missed doses, the ficlatuzumab will be discontinued permanently. However, if in the investigator's opinion there is evidence of clinical benefit, a subject with 2 consecutive missed doses may resume treatment after the AE has resolved to the minimum specifications in Table 4A or Table 4B. Contact the Sponsor-Investigator for consensus on subsequent treatment.

## 5.5.4 Treatment Interruption for Interstitial Lung Disease

In the event of acute onset (grade  $\geq$  2) or worsening pulmonary symptoms which are not thought to be related to underlying cancer, both cetuximab and ficlatuzumab should be interrupted and a prompt investigation of these symptoms should occur. Neither ficlatuzumab nor cetuximab retreatment should occur until these symptoms have resolved to grade 1. If interstitial lung disease is confirmed, both cetuximab and ficlatuzumab should be discontinued permanently and the patient should be treated appropriately.

## **5.5.5** Dose Modification for Hematologic Toxicity

While serious (Grade 3-4) myelosuppression has not been observed with ficlatuzumab monotherapy or the combination of ficlatuzumab with EGFR-inhibitors during phase I development, dose modifications are specified in <u>Table 4A</u> for neutropenia or thrombocytopenia, should either be observed during the course of this phase II study. As cetuximab does not cause myelosuppression, the cetuximab dose will not be affected by observed neutropenia or thrombocytopenia.

Table 4A. Ficlatuzumab and Cetuximab Dose Modifications for Hematologic Toxicity

| Adverse Event NCI CTCAE Toxicity Grade (CTCAE v. 4.0) | Ficlatuzumab Dose | Cetuximab Dose |
|---|---|---|
| Neutropenia | | |
| Grade 1-2<br>1 (1,500-1,999/mm³)<br>2 (1,000-1,499/mm³) | Maintain dose level | Maintain dose level |
| Grade ≥3:<br>3 (500-999/mm³)<br>4 (<500/mm³) | Hold dose. When recovered to Grade 2 or | Maintain dose level |

| | better, decrease by 1 dose level. | |
|---|---|---|
| Thrombocytopenia | | |
| Grade 1 (75,000/mm <sup>3</sup> -LLN) | Maintain dose level | Maintain dose level |
| Grade ≥ 2:<br>2 (50,000-74,999/mm³)<br>3 (25,000-49,999/mm³)<br>4 (<25,000/mm³) | Hold dose. Re-assess prior<br>to next scheduled dose.<br>When recovered to Grade<br>1 or better, decrease by 1<br>dose level. | Maintain dose level |

# 5.5.6 Dose Modification for Non-Hematologic Toxicity

Adverse events observed and deemed to be at least possibly related to study drug(s) will be managed according to the guidelines for dose interruption, delay, or reduction.

If the non-hematologic toxicity can be clearly and solely attributed to ficlatuzumab, the ficlatuzumab should be withheld or reduced as described below in <u>Table 4B</u>. If the non-hematologic toxicity is at least possibly related to both ficlatuzumab and cetuximab, then both study drugs should be modified as described below. If the non-hematologic toxicity can be clearly and solely attributed to cetuximab, the cetuximab should be withheld or reduced as described below in <u>Table 4B</u>.

Table 4B. Ficlatuzumab and Cetuximab Dose Reductions for Non-Hematologic Toxicity

| Adverse Event NCI CTCAE Toxicity Grade (CTCAE v. 4.0) | Ficlatuzumab Dose | Cetuximab Dose |
|---|---|---|
| Metabolic <sup>a</sup> Hypomagnesemia, Hypokalemia, Hypophosphatemia, or Hyponatremia | | |
| Grade ≥ 3, Asymptomatic | Administer PO or IV replacement and reassess. If Grade ≤2, continue drug at same dose level. (Same day re-assessment and dosing is permissible.) If AE does not recover to Grade ≤2, hold drug. | Administer PO or IV replacement and reassess. If Grade ≤2, continue drug at same dose level. (Same day re-assessment and dosing is permissible.) If AE does not recover to Grade ≤2, hold drug. |
| Grade ≥ 3, Symptomatic | Administer PO or IV replacement and reassess. If | Administer PO or IV replacement and reassess. If |

| Adverse Event | Ficlatuzumab Dose | Cetuximab Dose |
|---|---|---|
| NCI CTCAE Toxicity Grade | Ficiatuzumab Dose | Cetuximab Dose |
| (CTCAE v. 4.0) | | |
| , | ≤ Grade 2 <b>and</b> asymptomatic, | ≤ Grade 2 <b>and</b> |
| | then reduce by one dose | asymptomatic, then reduce |
| | level. (Same day re- | by one dose level. (Same day re-assessment and dosing is |
| | assessment and dosing is permissible.) If AE does not | permissible.) If AE does not |
| | recover to Grade ≤2 <b>and</b> | recover to Grade ≤2 <b>and</b> |
| | asymptomatic, hold drug. | asymptomatic, hold drug. |
| Hepatic Function | | |
| AST and/or ALT Elevation | | |
| Grade 2 | Reduce by one dose level | Reduce by one dose level |
| Grade ≥ 3 | Hold drug until ≤ grade 2 | Hold drug until ≤ grade 2 |
| 6.446 = 5 | then reduce by one dose level | then reduce by one dose<br>level |
| AST or ALT elevation >3x ULN and concomitant elevation of bilirubin >2x ULN | Discontinue ficlatuzumab | Discontinue cetuximab |
| Low Albumin | | |
| Grade 3 | No dose reduction | No dose reduction |
| Grade 4 | Reduce by one dose level | No dose reduction |
| <b>Edema:</b> Head/Facial/Neck edema and peripheral edema are to be managed individually. | | |
| Head/Facial/Neck Edema | | |
| <u>Tolerable</u> Grade ≤ 2 | No dose reduction. Treat with PO diuretics as clinically indicated. | No dose reduction |
| | Hold drug. <u>Administer</u><br><u>steroids <sup>c</sup></u> and/or PO or IV | No dose reduction |

| Adverse Event NCI CTCAE Toxicity Grade (CTCAE v. 4.0) | Ficlatuzumab Dose | Cetuximab Dose |
|---|---|---|
| Intolerable b Grade 2 (per opinion of treating investigator) or Grade ≥ 3 | diuretics as clinically indicated. Resume drug when ≤ tolerable grade 2 and reduce by one dose level. | |
| Peripheral Edema <u>Tolerable</u> Grade ≤ 2 | No dose reduction. Treat with PO diuretics as clinically indicated. | No dose reduction |
| Intolerable b Grade 2 (per the opinion of treating investigator) or Grade ≥ 3 | Hold drug. <u>Administer</u> <u>steroids of and/or PO or IV</u> diuretics as clinically indicated. Resume drug when ≤ <u>tolerable</u> grade 2 and reduce by one dose level. | No dose reduction |
| Fatigue | | |
| Grade ≥ 3, lasting more than 7 days | Hold drug until ≤ grade 2<br>then reduce by one dose level | Hold drug until ≤ grade 2<br>then reduce by one dose<br>level |
| Nausea/Vomiting | | |
| ≥ Grade 3 with maximal medical management | Hold drug until ≤ grade 2<br>then reduce by one dose level | Hold drug until ≤ grade 2<br>then reduce by one dose<br>level |
| Dermatologic events | | |

| Adverse Event NCI CTCAE Toxicity Grade (CTCAE v. 4.0) | Ficlatuzumab Dose | Cetuximab Dose |
|---|---|---|
| Rash, Acneiform<br>(Grade per <u>Table 5</u> below.) | | |
| ≥ Grade 3 | Maintain dose level | First Occurrence: Hold drug for two weeks. If improved to ≤ grade 2 then restart cetuximab at same dose level. If rash remains ≥ Grade 3 then discontinue cetuximab. |
| | | Second Occurrence: Hold drug for two weeks. If improved to ≤ grade 2 then restart cetuximab at dose level -1. If rash remains ≥ Grade 3 then discontinue cetuximab. |
| | | Third Occurrence: Hold drug for two weeks. If improved to ≤ grade 2 then restart cetuximab at dose level -2. If rash remains ≥ Grade 3 then discontinue cetuximab. |
| | | Fourth occurrence: discontinue cetuximab. |

| Adverse Event NCI CTCAE Toxicity Grade (CTCAE v. 4.0) | Ficlatuzumab Dose | Cetuximab Dose |
|---|---|---|
| Paronychia<br>(Grade per <u>Table 5</u> below.) | | |
| ≥ Grade 3 | Maintain dose level | First Occurrence: Hold drug for two weeks. If improved to ≤ grade 2 then restart cetuximab at same dose level. If paronychia remains ≥ Grade 3 then discontinue cetuximab. |
| | | Second Occurrence: Hold<br>drug for two weeks. If<br>improved to ≤ grade 2 then<br>restart cetuximab at dose<br>level -1. If paronychia<br>remains ≥ Grade 3 then<br>discontinue cetuximab. |
| | | Third Occurrence: Hold drug for two weeks. If improved to ≤ grade 2 then restart cetuximab at dose level -2. If paronychia remains ≥ Grade 3 then discontinue cetuximab. |
| | | Fourth occurrence: discontinue cetuximab. |
| <b>Pruritus</b> (Grade per <u>Table 5</u> below.) | | |
| ≥ Grade 3 | Maintain dose level | First Occurrence: Hold drug for two weeks. If improved to ≤ grade 2 then restart cetuximab at same dose level. If pruritus remains ≥ Grade 3 then discontinue cetuximab. |

| Adverse Event | Ficlatuzumab Dose | Cetuximab Dose |
|---|---|---|
| NCI CTCAE Toxicity Grade (CTCAE v. 4.0) | | |
| (CICAL V. 4.0) | | Second Occurrence: Hold drug for two weeks. If improved to ≤ grade 2 then restart cetuximab at dose level -1. If pruritus remains ≥ Grade 3 then discontinue cetuximab. |
| | | Third Occurrence: Hold drug for two weeks. If improved to ≤ grade 2 then restart cetuximab at dose level -2. If pruritus remains ≥ Grade 3 then discontinue cetuximab. |
| | | Fourth occurrence: discontinue cetuximab. |
| Rash, other<br>(Grade per <u>Table 5</u> below.) | | discontinue cetaximus. |
| ≥ Grade 3 | Maintain dose level | First Occurrence: Hold drug for two weeks. If improved to ≤ grade 2 then restart cetuximab at same dose level. If rash remains ≥ Grade 3 then discontinue cetuximab. |
| | | Second Occurrence: Hold drug for two weeks. If improved to ≤ grade 2 then restart cetuximab at dose level -1. If rash remains ≥ Grade 3 then discontinue cetuximab. |
| | | Third Occurrence: Hold drug<br>for two weeks. If improved to<br>≤ grade 2 then restart<br>cetuximab at dose level -2. If |

| Adverse Event NCI CTCAE Toxicity Grade (CTCAE v. 4.0) | Ficlatuzumab Dose | Cetuximab Dose |
|---|---|---|
| | | rash remains ≥ Grade 3 then discontinue cetuximab. |
| | | Fourth occurrence: discontinue cetuximab. |
| Other, Grade ≥ 3 Events at least possibly related to ONLY ficlatuzumab | Hold drug until ≤ grade 1 or baseline, then reduce by one dose level. | Maintain dose level. |
| Other, Grade ≥ 3 Events at least possibly related to ONLY cetuximab | Maintain dose level. | Hold drug until ≤ grade 1 or baseline, then reduce by one dose level. |
| Other, Grade ≥ 3 Events at least possibly related to both ficlatuzumab and cetuximab | Hold drug until ≤ grade 1 or baseline, then reduce by one dose level. | Hold drug until ≤ grade 1 or baseline, then reduce by one dose level. |
| Other, Grade ≥ 3 Events that are NOT related to or expected from either ficlatuzumab or cetuximab | If determined to be clinically significant, in the judgement of the treating investigator, hold until resolved to ≤ grade 1 or baseline and restart at same dose. | |

- a. Sustained deficiency may require both chronic oral **and** IV replacement. An EKG is strongly recommended in the event of: 1) symptomatic Grade ≥ 3 hypomagnesemia or hypokalemia or 2) asymptomatic Grade 4 hypomagnesemia or hypokalemia. Interventions, including hospitalization as necessary for correction of electrolyte derangement, should occur in accordance with clinical severity and investigator judgment.
- b. "Intolerable" is to be determined by treating investigator opinion.
- C. Suggested steroid pulse of Prednisone 40 mg/daily for 5 days.

#### **5.5.7 Dermatologic Toxicity**

Cetuximab-related dermatologic toxicity should be graded according to the criteria outlined in Table 5 below. According to physician judgment, if a patient experiences ≥ grade 3 rash, cetuximab treatment adjustments should be made according to <u>Table 4B</u> above. In patients with mild and moderate skin adverse events, cetuximab should continue without adjustment.

**Table 5: Grading of Cetuximab-Related Skin Changes** 

| | 1 | 2 | 3 | 4 |
|---|---|---|---|---|
| Pruritus* | Mild or localized | Intense or<br>widespread | Intense or<br>widespread and<br>interfering with<br>ADL | - |
| Rash/acneiform* | Papules and/or pustules covering <10% BSA, which may or may not be associated with symptoms of pruritus or tenderness | Papules and/or pustules covering 10-30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; associated with psychosocial impact; limiting instrumental ADLI; Responds promptly to symptomatic treatment | Papules and/or pustules covering > 30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; limiting self-care ADL; associated with local superinfection with oral antibiotics indicated; Prolonged. | Papules and/or pustules covering any % BSA, which may or may not be associated with symptoms of pruritus or tenderness and are associated with extensive superinfection with IV antibiotics indicated; life threatening consequences |
| Paronychia Onset of grade 3 will require dose modification for cetuximab. See Table 4B above. | Nail fold edema<br>or erythema;<br>disruption of the<br>cuticle | Localized intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, antiviral); nail fold edema or erythema with pain; associated with discharge or nail plate separation; limiting instrumental ADL | Surgical<br>intervention or IV<br>antibiotics<br>indicated; limiting<br>self<br>care ADL | - |
## **Cetuximab-Related Rash Management**

Skin rash, ranging from dry skin and erythema to a pustular eruption is extremely common during cetuximab therapy. Biopsy of the papulopustular rash demonstrates histopathologic suppurative inflammation and not acne vulgaris. Although the initial rash is sterile, superinfection may occur.

Patients developing dermatologic AEs while receiving cetuximab should be monitored for the development of inflammatory or infectious sequelae, and appropriate treatment of these symptoms initiated. Below are suggestions for managing cetuximab-induced rash, adapted from the NCCN Task Force for the Management of Dermatologic Toxicities Associated with EGFR Inhibition in Patients with Cancer.47 In the event of severe rash not responsive to topical treatments or oral antibiotics, dose modification per Table 4B is indicated.

- Moisturizers: Use of topical emollients to prevent and alleviate skin dryness is strongly advised. Examples include Aquaphor Ointment, Cetaphil Cream, Neutrogena Norwegian Formula Hand Cream, and Vaseline Intensive Care Advanced Healing Lotion.
- **Soap:** A mild, neutral pH soap is recommended.
- Antibiotics: Topical clindamycin or erythromycin, or an oral tetracycline family antibiotic
  (e.g. tetracycline, minocycline, doxycycline) should be considered in the case of
  superinfection or suspected superinfection. Oral minocycline, tetracycline or doxycycline
  may be given prophylactically to patients with a history of severe acneiform eruption
  during prior cetuximab therapy.
- **Antihistamines**: Diphenhydramine or hydroxyzine may be helpful to control itching.
- **Topical Steroids**: Topical therapy with a low potency steroid to the face (e.g. hydrocortisone valerate 0.2%) or a mid-potency steroid to the body (e.g. triamcinolone acetonide 0.1%) may be used for management of cetuximab rash.
- **Sunlight**: It is recommended that patients wear sunscreen (at least SPF 40) and hats and limit sun exposure while receiving cetuximab as sunlight can exacerbate any skin reactions that may occur.
- Over-the-counter medications: Over-the-counter acne vulgaris medications (e.g. benzoyl peroxide) are not advised.
- Retinoids: Use is not advised.

#### 5.5.8 Cetuximab Infusion Reaction

A cetuximab infusion reaction will be managed as described in <u>Table 6</u> below. If there is any question as to whether an observed reaction is an infusion reaction of Grades 1-4, Dr. Julie Bauman should be contacted immediately to discuss and grade the reaction.

Should an infusion reaction occur, retreatment will be managed as follows: Once a cetuximab infusion rate has been decreased due to an infusion reaction, it will remain decreased for all subsequent infusions. If the subject has a second infusion reaction with the slower infusion rate, the infusion should be stopped, and the subject should receive no further cetuximab treatment. If a subject that experienced an initial cetuximab infusion reaction experiences a Grade 3 or 4 infusion reaction at any time, the subject should receive no further cetuximab treatment.

**Table 6: Management of Cetuximab Infusion Reaction** 

| Grade | Management |
|---|---|
| Grade 1: Transient flushing or rash; drug fever < 38° C (< 100.4° F) | For mild infusion reactions manifesting only as delayed drug fever, consider administering prophylactic antihistamine medications for subsequent doses. Maintain the cetuximab dose but slow the infusion rate by 50%. Acetaminophen or a non-steroidal anti-inflammatory drug (NSAID) may be administered prior to subsequent cetuximab infusions, if not otherwise contraindicated in subjects. |
| Grade 2: Rash; flushing; urticaria; dyspnea; drug fever ≥ 38° C (≥ 100.4° F) | For moderate infusion reactions manifesting only as delayed drug fever, slow the infusion rate for cetuximab by 50%, and consider administration of antihistamine medications and/or steroidal medications. Maintain the cetuximab dose. Acetaminophen or a non-steroidal anti-inflammatory drug (NSAID) may be administered prior to subsequent cetuximab infusions, if not otherwise contraindicated in subjects. |
| Grade 3: Symptomatic bronchospasm with or without urticaria; parenteral medication(s) indicated; allergy- related edema/angioedema; hypotension | Severe infusion reactions requires immediate interruption of cetuximab infusion and permanent discontinuation from further treatment with cetuximab. Appropriate medical therapy including epinephrine, corticosteroids, diphenhydramine, bronchodilators, and oxygen should be available for use in the treatment of such reactions. Subjects should be carefully observed until the complete resolution of all signs and symptoms. |

| Grade 4: | NO FURTHER CETUXIMAB |
|---|---|
| Anaphylaxis | Life-threatening infusion reactions require immediate interruption of cetuximab infusion and permanent discontinuation from further treatment with cetuximab. Appropriate medical therapy including |
| | epinephrine, corticosteroids, diphenhydramine, bronchodilators, and oxygen should be available for use in the treatment of such reactions. Subjects should be carefully observed until the complete resolution of all signs and symptoms. |

#### 6. RESPONSE ASSESSMENT

Patients are to be re-evaluated for response every 8 weeks, +/- 7 days during at least Cycle 1 through Cycle 12. Disease assessment is performed per standard of care and per physician's determination of clinical indication.

Consistent with standard of care, subjects who remain on treatment after cycle 12 can be transitioned to re-evaluation for response every 12 weeks, +/- 14 days. Refer to Section 8.3.3.

Response and progression will be evaluated in this study using the international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1).<sup>48</sup> Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used.

The objective malignant disease evaluation will determine the subject's response, except when the subject presents with symptomatic deterioration ("clinical progression"). Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time should be classified as having *symptomatic deterioration*.

## **6.1 Malignant Disease Evaluation**

To assess objective response, it is necessary to estimate the overall tumor burden at baseline to which subsequent measurements will be compared. Measurable disease is defined by the presence of at least one measurable lesion.

All measurements should be recorded in metric notation by use of a ruler or calipers. The same method of assessment and the same technique should be used to characterize each identified lesion at baseline and during follow-up. All baseline evaluations should be performed as closely as possible to the beginning of treatment and never more than 28 days before registration.

Refer to <u>Section 8.1</u> Screening/Pre-treatment Evaluations.

The term unevaluable in reference to measurability will not be used because it does not provide additional meaning or accuracy.

At baseline, the primary tumor and pathologic neck lymph nodes will be characterized as either measurable or non-measurable.

#### 6.1.1 Measurable Disease

Primary and/or Metastatic HNSCC Tumors (non-Lymph node):

• Lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm (2.0 cm) with conventional techniques or as ≥ 10 mm (1.0 cm) with spiral CT scan.

#### Lymph Nodes:

- Lymph nodes are considered pathologic and measurable if short axis ≥ 15 mm.
- Lymph nodes are considered pathologic but non-measurable if short axis ≥ 10 mm but <</li>
   15 mm.
- Lymph nodes are considered non-pathologic and non-measurable if short axis < 10 mm.

#### 6.1.2 Non-measurable disease

All other lesions, including small lesions [longest diameter < 20 mm (2.0 cm) with conventional techniques or < 10 mm (1.0 cm) with spiral CT scan] are truly non-measurable lesions.

Lesions considered to be truly non-measurable include the following: bone lesions, leptomeningeal disease, ascites, pleural/pericardial effusion, inflammatory breast disease, lymphangitis cutis/pulmonis, abdominal masses that are not confirmed and followed by imaging techniques, and cystic lesions.

#### 6.1.3 Target Lesions

Measurable lesions up to a maximum of 2 lesions per organ and 5 lesions in total, representative of all involved organs, should be identified as target lesions and recorded and measured at baseline. Target lesions should be selected on the basis of their size (lesions with the longest diameter), be representative of all involved organs, but in addition should be those that lend themselves to reproducible repeated measurements. It may be the case that, on occasion, the largest lesion does not lend itself to reproducible measurement in which circumstance the next largest lesion which can be measured reproducibly should be selected. A sum of the diameters (longest for non-nodal lesions, short axis for nodal lesions) for all target lesions will be calculated and reported as the baseline sum diameters. If lymph nodes are to be included in the

sum, then only the short axis is added into the sum. The baseline sum diameters will be used as reference to further characterize any objective tumor regression in the measurable dimension of the disease.

## 6.1.4 Non-target Lesions

All other lesions (or sites of disease) including any measurable lesions over and above the 5 target lesions should be identified as non-target lesions and should also be recorded at baseline. Measurements of these lesions are not required, but the presence, absence, or in rare cases unequivocal progression of each should be noted throughout follow-up.

## **6.2 Response Criteria**

## 6.2.1 Evaluation of Target Lesions

## **Complete Response (CR) of Target Lesions**

Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.

#### Partial Response (PR) of Target Lesions

At least a 30% decrease in the sum of target lesion diameters (longest diameter of non-nodal lesions; short axis diameter of the target lymph nodes), taking as reference the *baseline sum diameter*.

#### **Stable Disease (SD) of Target Lesions**

Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.

#### **Progressive Disease (PD) of Target Lesions**

At least a 20% increase in the sum of target lesion diameters (longest diameter of non-nodal lesions; short axis diameter of the target lymph nodes), taking as reference the *smallest sum diameter* recorded since the baseline sum diameter measurements. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Note: the appearance of one or more new lesions is also considered progressions.

## **6.2.2 Evaluation of Non-target Lesions**

All other lesions or sites of disease. Measurements of these lesions are not required, but the presence, absence, stable, or progression of each must be noted throughout follow-up.

#### **Complete Response (CR) of Non-target Lesions**

The disappearance of all nontarget lesions.

#### Partial Response/Stable Disease (SD) of Non-target Lesions

Confidential

 v10, 05/23/2023

The persistence of one or more nontarget lesion(s).

## **Progressive Disease (PD) of Non-target Lesions**

The appearance of one or more new lesions and/or unequivocal progression of existing nontarget lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.

Although a clear progression of "non-target" lesions only is exceptional, the opinion of the treating physician should prevail in such circumstances, and the progression status should be confirmed at a later time by the review panel (or Principal Investigator).

## **Evaluation of Patient's Best Overall Response**

The best overall response is the best response recorded from registration until disease progression/recurrence, taking as reference for progressive disease the smallest measurements recorded since registration. <u>Table 7</u> below provides overall responses for all possible combinations of tumor responses in target and nontarget lesions, with or without new lesions.

To be assigned a status of stable disease, measurements must have met the stable disease criteria at least once after study entry at a minimum interval of eight weeks (+/- 1 week).

| Target | Non-Target Lesions | New | Overall | Best Overall F |
|---------|--------------------|---------|----------|----------------|
| Lesions | | Lesions | Response | when Confirr |

Table 7: Evaluation for Patients with Measurable Disease (i.e., Target Disease)

| Target<br>Lesions | Non-Target Lesions | New<br>Lesions | Overall<br>Response | Best Overall Response<br>when Confirmation is<br>Required* |
|---|---|---|---|---|
| CR | CR | No | CR | ≥4 wks. Confirmation** |
| CR | Non-CR/Non-PD | No | PR | |
| CR | Not evaluated | No | PR | >4 wks. Confirmation** |
| PR | Non-CR/Non-PD/not evaluated | No | PR | |
| SD | Non-CR/Non-PD/not evaluated | No | SD | Documented at least once<br>>4 wks. from baseline** |
| PD | Any | Yes or No | PD | |
| Any | PD*** | Yes or No | PD | No prior SD, PR or CR |
| Any | Any | Yes | PD | |

<sup>\*</sup> See RECIST 1.1 manuscript for further details on what is evidence of a new lesion.

Note: Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time should be reported as "symptomatic

<sup>\*\*</sup> Only for non-randomized trials with response as primary endpoint.

<sup>\*\*\*</sup> In exceptional circumstances, unequivocal progression in non-target lesions may be accepted as disease progression.

deterioration." Every effort should be made to document the objective progression even after discontinuation of treatment.

CR = complete response; PR = partial response; SD = stable disease; PD = progressive disease

## **First Documentation of Response**

The time between initiation of therapy and first documentation of PR or CR.

## **Confirmation of Response**

To be assigned a status of complete or partial response, changes in tumor measurements must be confirmed by repeat assessments performed no less than four weeks after the criteria for response are first met.

## **Duration of Response**

Duration of overall response - the period measured from the time that measurement criteria are met for complete or partial response (whichever status is recorded first) until the first date that recurrent or progressive disease is objectively documented, taking as reference the smallest measurements recorded since treatment started.

## **Duration of Overall Complete Response**

The period measured from the time measurement criteria are met for complete response until the first date that recurrent disease is objectively documented.

#### **Duration of Stable Disease**

A measurement from registration until the criteria for disease progression is met, taking as reference the smallest measurements recorded since registration. To be assigned a status of stable disease, measurements must have met the stable disease criteria at least once after study entry at a minimum interval of eight weeks (+/- 1 week).

#### Survival

Survival will be measured from the date of entry on study.

## Time to Progression and Progression-free survival

This interval will be measured from the date of entry on the study to the appearance of new metastatic lesions or objective tumor progression.

Progression-free survival (PFS) will be calculated from treatment initiation to disease progression or death from any cause.

#### 6.3 Methods of Measurement

Disease assessment is performed per standard of care.

All measurements should be taken and recorded in metric notation using a ruler or calipers. All baseline evaluations should be performed as closely as possible to the beginning of treatment and never more than 28 days before registration.

The same method of assessment and the same technique should be used to characterize each identified and reported lesion at baseline and during follow-up. Imaging-based evaluation is preferred to evaluation by clinical examination unless the lesion(s) being followed cannot be imaged but are assessable by clinical exam and measureable by ruler or caliper (clinical lesions).

Diagnostic CT scan is the preferred modality.

MRI may be substituted per investigator judgment (e.g., MRI of the neck with contrast, in cases where patient has an iodinated contrast allergy despite premedication).

PET/CT may only be used for tumor measurements if the CT component is of diagnostic quality. PET/CT where CT is performed only for attenuation correction is not of sufficient quality for RECIST measurements.

<u>Clinical lesions</u> Clinical lesions will only be considered measurable when they are superficial (e.g., skin nodules and palpable lymph nodes) and ≥10 mm diameter as assessed using a ruler or calipers (e.g., skin nodules). In the case of skin lesions, documentation by color photography, including a ruler to estimate the size of the lesion, is recommended.

<u>Conventional CT and MRI</u> This guideline has defined measurability of lesions on CT scan based on the assumption that CT slice thickness is 5 mm or less. If CT scans have slice thickness greater than 5 mm, the minimum size for a measurable lesion should be twice the slice thickness. MRI is also acceptable in certain situations (e.g. for body scans).

Use of MRI remains a complex issue. MRI has excellent contrast, spatial, and temporal resolution; however, there are many image acquisition variables involved in MRI, which greatly impact image quality, lesion conspicuity, and measurement. Furthermore, the availability of MRI is variable globally. As with CT, if an MRI is performed, the technical specifications of the scanning sequences used should be optimized for the evaluation of the type and site of disease. Furthermore, as with CT, the modality used at follow-up should be the same as was used at baseline and the lesions should be measured/assessed on the same pulse sequence. It is beyond the scope of the RECIST guidelines to prescribe specific MRI pulse sequence parameters for all scanners, body parts, and diseases. Ideally, the same type of scanner should be used and the image acquisition protocol should be followed as closely as possible to prior scans. Body scans

should be performed with breath-hold scanning techniques, if possible.

<u>PET-CT</u> At present, the low dose or attenuation correction CT portion of a combined PET-CT is not always of optimal diagnostic CT quality for use with RECIST measurements. However, if the site can document that the CT performed as part of a PET-CT is of identical diagnostic quality to a diagnostic CT (with IV and oral contrast), then the CT portion of the PET-CT can be used for RECIST measurements and can be used interchangeably with conventional CT in accurately measuring cancer lesions over time. Note, however, that the PET portion of the CT introduces additional data which may bias an investigator if it is not routinely or serially performed.

<u>Ultrasound</u> Ultrasound is not useful in assessment of lesion size and should not be used as a method of measurement. Ultrasound examinations cannot be reproduced in their entirety for independent review at a later date and, because they are operator dependent, it cannot be guaranteed that the same technique and measurements will be taken from one assessment to the next. If new lesions are identified by ultrasound in the course of the study, confirmation by CT or MRI is advised. If there is concern about radiation exposure at CT, MRI may be used instead of CT in selected instances.

<u>Endoscopy</u>, <u>Laparoscopy</u> The utilization of these techniques for objective tumor evaluation is not advised. However, such techniques may be useful to confirm complete pathological response when biopsies are obtained or to determine relapse in trials where recurrence following complete response (CR) or surgical resection is an endpoint.

<u>Cytology</u>, <u>Histology</u> These techniques can be used to differentiate between partial responses (PR) and complete responses (CR) in rare cases (e.g., residual lesions in tumor types, such as germ cell tumors, where known residual benign tumors can remain).

The cytological confirmation of the neoplastic origin of any effusion that appears or worsens during treatment when the measurable tumor has met criteria for response or stable disease is mandatory to differentiate between response or stable disease (an effusion may be a side effect of the treatment) and progressive disease.

<u>FDG-PET</u> While FDG-PET response assessments need additional study, it is sometimes reasonable to incorporate the use of FDG-PET scanning to complement CT scanning in assessment of progression (particularly possible 'new' disease). New lesions on the basis of FDG-PET imaging can be identified according to the following algorithm:

• Negative FDG-PET at baseline, with a positive FDG-PET at follow-up is a sign of PD based on a new lesion.

- No FDG-PET at baseline and a positive FDG-PET at follow-up: If the positive FDG-PET at follow-up corresponds to a new site of disease confirmed by CT, this is PD. If the positive FDG-PET at follow-up is not confirmed as a new site of disease on CT, additional follow-up CT scans are needed to determine if there is truly progression occurring at that site (if so, the date of PD will be the date of the initial abnormal FDG-PET scan). If the positive FDG-PET at follow-up corresponds to a pre-existing site of disease on CT that is not progressing on the basis of the anatomic images, this is not PD.
- FDG-PET may be used to upgrade a response to a CR in a manner similar to a biopsy in cases where a residual radiographic abnormality is thought to represent fibrosis or scarring. The use of FDG-PET in this circumstance should be prospectively described in the protocol and supported by disease-specific medical literature for the indication. However, it must be acknowledged that both approaches may lead to false positive CR due to limitations of FDG-PET and biopsy resolution/sensitivity.

Note: A 'positive' FDG-PET scan lesion means one which is FDG avid with an uptake greater than twice that of the surrounding tissue on the attenuation corrected image.

#### 7. DRUG INFORMATION

#### 7.1 Ficlatuzumab

## 7.1.1 Study Drug Materials

The Aveo Pharmacy Manual should be referenced for drug preparation and administration information.

Ficlatuzumab Concentrate for Injection, 50 mg/mL, is formulated in 10 mM histidine buffer pH 5.8. The formulation also includes 142 mM arginine (for isotonicity) and 0.01% polysorbate-80. The product is sterile filtered and aseptically filled into washed and depyrogenated 4-mL and 20 mL glass vials. An excess fill is provided in the vial to ensure that the label fill of 4.0 mL can be withdrawn. The product is a clear to slightly opalescent, colorless to slightly yellow, solution.

Ficiatuzumab Concentrate for Injection is to be administered by IV infusion as an admixture with normal saline solution. The admixture solution in an IV bag is connected to an infusion set containing a 0.22  $\mu$ m low protein-binding in-line filter. The IV bag and the infusion set containing the in-line filter have been shown to be compatible with the admixture. The filtered admixture solution is clear to slightly opalescent.

## 7.1.2 Ficlatuzumab Study Drug Storage

Ficiatuzumab is to be stored under refrigerated conditions ( $2^{\circ}$  C -  $8^{\circ}$ C) and in a secure location.

Note: No other use of ficlatuzumab study drug intended for use in this trial is authorized by the

sponsor. The investigator (or designee) will be responsible for the appropriate handling and disposition of residual study drug in partially used vials.

Vial Labels: Ficlatuzumab vial labels will bear the appropriate label text for investigational agents, as required by governing regulatory agencies.

Complete study drug information (including packaging, labeling, storage and disposition) is provided in the Ficlatuzumab Investigator's Brochure (IB).

## 7.1.3 Study Drug Accountability

The local Investigator will be responsible for the supplied study drug, its administration, and accountability. The investigational product must only be used for this protocol and must be stored and accounted for consistent with regulatory requirements, the Aveo Pharmacy Manual, and this protocol. An accurate record of all study drugs received, dispensed, returned, and destroyed must be maintained.

#### 7.2 Cetuximab

Refer to the package insert for additional information.

<u>Formulation</u>: Cetuximab is an anti-EGFR receptor humanized chimeric monoclonal antibody. Cetuximab is expressed in SP2/0 myeloma cell line, grown in large scale cell culture bioreactors, and purified to a high level purity using several purification steps including protein A chromatography, ion exchange chromatography, low pH treatment, and nanofiltration. Cetuximab is not known to be a vesicant.

<u>Safety Precautions</u>: Appropriate mask, protective clothing, eye protection, gloves and Class II vertical-laminar-airflow safety cabinets are recommended during preparation and handling.

<u>Preparation and Administration</u>: Cetuximab must not be administered as an IV push or bolus. Cetuximab must be administered with the use of a low protein binding 0.22-micrometer in-line filter.

Cetuximab is supplied as a 50-mL, single-use vial containing 100 mg of cetuximab at a concentration of 2 mg/mL in phosphate buffered saline. The solution should be clear and colorless and may contain a small amount of easily visible white amorphous cetuximab particulates. DO NOT SHAKE OR DILUTE.

Cetuximab can be administered via infusion pump or syringe pump.

#### Infusion Pump:

1. Draw up the volume of a vial using a sterile syringe attached to an appropriate needle (a vented spike or other appropriate transfer device may be used).

- 2. Fill cetuximab into a sterile evacuated container or bag such as glass containers, polyolefin bags (eg, Baxter Intravia), ethylene vinyl acetate bags (eg, Baxter Clintec), DEHP plasticized PVC bags (eg, Abbott Lifecare), or PVC bags.
- 3. Repeat procedure until the calculated volume has been put in to the container. Use a new needle for each vial.
- 4. Administration must be through a low protein binding 0.22-micrometer in-line filter (placed as proximal to the patient as practical).
- 5. Affix the infusion line and prime it with cetuximab before starting the infusion.
- 6. Maximum infusion rate should not exceed 5 mL/min (10 mg/min).
- 7. Use 0.9% saline solution to flush line at the end of infusion.

## Syringe Pump:

- 1. Draw up the volume of a vial using a sterile syringe attached to an appropriate needle (a vented spike may be used).
- 2. Place the syringe into the syringe driver of a syringe pump and set the rate.
- 3. Administration must be through a low protein binding 0.22-micrometer in-line filter rated for syringe pump use (placed as proximal to the patient as practical).
- 4. Connect up the infusion line and start the infusion after priming the line with cetuximab.
- 5. Repeat procedure until the calculated volume has been infused.
- 6. Use a new needle and filter for each vial.
- 7. Maximum infusion rate should not exceed 5 mL/min (10 mg/min).
- 8. Use 0.9% saline solution to flush line at the end of infusion.

Cetuximab should be piggybacked to the patient's infusion line.

Following the cetuximab infusion, a one-hour observation period is recommended.

#### Storage Requirements/Stability

Store vials under refrigeration at 2° C to 8° C (36° F to 46° F). DO NOT FREEZE. Increased particulate formation may occur at temperatures at or below 0°C. This product contains no preservatives. Preparations of cetuximab in infusion containers are chemically and physically stable for up to 12 hours at 2° C to 8° C (36° F to 46° F) and up to 8 hours at

v10, 05/23/2023

controlled room temperature (20° C to 25° C; 68° F to 77° F). Discard any remaining solution in the infusion container after 8 hours at controlled room temperature or after 12 hours at 2° to 8° C. Discard any unused portion of the vial.

#### Supply

Cetuximab is commercially available in the U.S.

## 8. STUDY PROCEDURES/EVALUATIONS

Schedule of Assessments. See Appendix C for Study Calendar.

#### Coronavirus/COVID-19 Considerations

As of March 2020, special considerations were implemented in the conduct of clinical trials during the COVID-19 public health emergency. Investigators must determine if changes are needed prior to IRB approval in order to eliminate apparent immediate hazard as allowed by regulations. The safety of subjects and others is priority, and the integrity of the study/study data must also be considered. Any changes/deviations related to the COVID-19 pandemic must be clearly documented as such and particular attention made to account for any missing data.

Should an in-person visit not be feasible or present immediate hazard to the subject, a phone contact should be performed to assess adverse events, concomitant medications, and ECOG performance status, as applicable for the specific visit. Additionally, the study questionnaires, Tobacco Use Assessment and FACT-H&N, can be done by phone or other method as appropriate.

Other potential changes and specific situations can be discussed with the Sponsor-Investigator as applicable/needed.

## 8.1 Screening/Pre-treatment evaluations

NOTE: All baseline evaluations should be performed as closely as possible to the beginning of treatment but <u>must</u> be performed within 28 days prior to registration unless otherwise indicated.

Written informed consent (prior to screening procedures)

- History and physical examination, including vital signs, weight, height, and ECOG performance status determination
- Documentation of medications subject is currently taking
- Complete blood count, including platelets, and differential
- Blood chemistry studies:
  - o BUN, creatinine, electrolytes (K<sup>+</sup>, Na<sup>+</sup>, Cl<sup>-</sup>, CO<sub>2</sub>), glucose, calcium, magnesium
    - Note: Patients may be supplemented to achieve acceptable electrolyte values
- Liver function tests:
  - Total protein, albumin, total bilirubin, AST (SGOT), ALT (SGPT), and alkaline phosphatase
- Documentation of calculation of corrected calcium for eligibility criterion
- For women of child bearing potential: Urine pregnancy test within <u>14 days</u> prior to registration to rule out pregnancy. (Note, negative pregnancy test must be confirmed again within 3 days prior to first study treatment.)
- Baseline tumor measurements within 28 days prior to registration.
- For oropharyngeal cases and unknown primary: HPV status (p16) status must be known or established and recorded at baseline (randomization is stratified by HPV status and documentation must be sent with the registration; see <u>Section 4</u>).
- Tobacco history assessment form (See Appendix D) (may be performed at screening or prior to study treatment on day 1; the assessment can be performed by method other than in-person, if needed, and the method used must be documented)
- Quality of life assessment (FACT-H&N Symptom Index) (may be performed at screening or prior to study treatment on day 1; the assessment can be performed by method other than in-person, if needed, and the method used must be documented)
- Research blood samples for correlative studies (may be performed at screening or prior to study treatment on day 1)
- Research biopsy of tumor tissue before first study drug administration (See <u>Section</u>
   9.2 for more information.)
- Confirm archived tumor specimens prior to cetuximab exposure are available for correlative research as outlined in <u>Section 9.1</u>. (Note: This is not an eligibility requirement and subjects can be randomized without this confirmation.)

#### 8.2 Registration & Randomization

Once deemed eligible, subject registration will be emailed to the sponsor. The randomization assignment will be returned to the site via email, typically within the day, or the following day

(including weekends).

## 8.3 Evaluations during study treatment

## 8.3.1 Every Two Weeks – Day 1 and Day 15 of each cycle (+/- 3 days)

**Note**: The following may be performed on the day of or within the 3 days prior to study drug administration. If the subject is deemed not acceptable for drug administration, refer to the visit delay and skipped visit description in <u>Section 5.5</u>. Subjects can return within the +3-day window, in 1 week, or for the next regularly scheduled treatment. If appropriate, the visit can be skipped and treatment can occur on schedule with the next regularly scheduled treatment (i.e., 2 weeks later).

- Physical examination, including vital signs, weight and ECOG performance status
- Adverse Event/Toxicity assessment with attribution
- Update of concomitant medications
- Complete blood count, including platelets and differential
- Blood chemistries:
  - o BUN, creatinine, electrolytes (K<sup>+</sup>, Na<sup>+</sup>, Cl<sup>-</sup>, CO<sub>2</sub>), glucose, calcium, magnesium
    - Note: Refer to <u>Table 4B</u> regarding grading, repletion, holding treatment, and/or dose reductions.
- Liver function tests:
  - o total protein, albumin, total bilirubin, AST (SGOT), ALT (SGPT), and alkaline phosphatase
- Study drug administration
  - o For both agents: Recalculate the doses of both ficiatuzumab and cetuximab only if there is a ≥ 10% change in weight. Exception: If, in the opinion of the treating investigator, weight change of ≥ 10% is due to edema, recalculation of the ficiatuzumab dose is not required. This decision must be clearly documented.

# 8.3.2 Every 8 Weeks (the end of even cycles – "Day 28"/8 weeks, 16 weeks, etc.)

- Quality of life assessment (FACT-H&N) end of cycle 2 and cycle 6 only.
  - The FACT-H&N may be done cycle 3, day 1/cycle 7, day 1 for subjects who remain on treatment.
  - If a subject stops treatment per the cycle 2 or cycle 6 scan, the FACT-H&N scheduled for C2D28 or C6D28 can be done at the End of Treatment visit.

- Tumor measurements according to RECIST 1.1 may be done during the last week of an even cycle, by CT scan or MRI.
  - Tumor measurements must be performed every 8 weeks, +/- 7 days for (at least) the first 12 cycles. (See <u>Section 8.3.3</u> regarding an optional tumor measurements schedule for subjects on treatment longer than 12 cycles.)
  - The schedule is independent of any treatment delays within the 2 cycles since the prior response assessment. (See <u>Section 5.5.1</u> regarding missed and/or skipped visits.)
  - The Response Assessment must be completed prior to drug administration at day
     1 of the following cycle.
- Research blood samples for correlative studies (these may be drawn simultaneously
  with the pre-treatment labs for the following cycle).

# 8.3.3 OPTIONAL: Every 12 Weeks Cycle 13+ ("Day 28" of every 3<sup>rd</sup> cycle after Cycle 12)

Tumor assessments for this trial are performed per standard of care. This optional transition to an every-12-week assessment is consistent with standard of care. This transition is **optional** and can occur **only if** it is appropriate as assessed on a patient-by-patient basis.

Transition to every-12-week tumor assessment will not affect the every-2-week drug administration treatment plan described in <u>Section 5</u> of this protocol.

- Subjects who remain on treatment past Cycle 12 (Cycle 13+) can be transitioned from every-8-week (+/- 7 days) tumor assessment to every-12-week (+/- 14 days) tumor assessment.
  - For example, a subject who has stable disease, partial response, or complete response per the Cycle 12, Day 28 scan can have their next scan performed on Cycle 15, Day 28, then Cycle 18, Day 28, Cycle 21, Day 28, and so forth.
  - The tumor assessment will be scheduled for Day 28 of every 3<sup>rd</sup> cycle (+/- 14 days).
  - The schedule is independent of any treatment delays within the 3 cycles since the prior assessment. (See <u>Section 5.5.1</u> regarding missed and/or skipped visits.)
  - The Response Assessment must be completed prior to drug administration on day 1 of the following cycle.
- Research blood samples for correlative studies will be drawn (blood may be drawn simultaneously with the pre-treatment labs for the following cycle).

#### 8.4 End-of-treatment (EOT) evaluations

- Patients who discontinue treatment for any reason will have an evaluation with the
  following tests, if possible <u>unless performed within the previous 2 weeks</u> (except as
  noted below) and unless otherwise indicated below. The EOT evaluations should be
  performed as soon as possible but within 30 days after the **off-treatment decision**date.
- Physical examination, including vital signs, weight and ECOG performance status
- Adverse Event/Toxicity assessment with attribution
- Update of concomitant medications
- Complete blood count, including platelets and differential
- Blood chemistries:
  - o BUN, creatinine, electrolytes (K<sup>+</sup>, Na<sup>+</sup>, Cl<sup>-</sup>, CO<sub>2</sub>), glucose, calcium, magnesium
- Liver function tests:
  - Total protein, albumin, total bilirubin, AST (SGOT), ALT (SGPT), and alkaline phosphatase
- Research blood for correlative studies
- For subjects that end treatment at C2D28 or C6D28, Quality of life (QoL) assessment (FACT-H&N)
  - Subjects that end treatment after C4D28 but prior to C6D28 due to expiration of the study drug will complete the QoL assessment at the EOT visit
- Tumor measurements according to RECIST 1.1 (<u>unless performed within the previous</u>
   28 days if it is an appropriate standard of care procedure the EOT tumor
   measurement will not be performed only for the research)

## 8.5 Post-treatment follow-up

#### 8.5.1 Adverse Event and Concomitant Medication Follow-up

AEs and SAEs will be followed per the details below regardless of the reason the subject ended treatment.

- Subjects will be followed for AEs (including SAEs) and pregnancy for at least 60 days after last dose of study drug(s) or until the initiation of subsequent antineoplastic therapy, whichever is earlier.
- Only new AEs that are considered related to the drug and pregnancy need to be documented during the 60 days.

- Any of related AEs that are SAEs must be reported as an SAE to the sponsor.
- AEs that are determined to be related to the study drug, whether documented during treatment or during follow-up, will be followed until resolution or stabilization.
- New concomitant medications do not need to be documented.

If a subject starts any new antineoplastic therapy, collection and follow up of AEs will stop, including AEs considered related/possibly related to the study drug, but SAEs that are considered related/possibly related may require continued assessment. Contact the Sponsor-Investigator for guidance.

## 8.5.2 Discontinuation of treatment WITHOUT progressive disease

If a patient discontinues treatment **without** progressive disease (clinical progression or radiologically assessed progression), he/she will be followed every 8 weeks (+/- 2 weeks) until progression of disease.

- AE/SAE assessment, per <u>Section 8.5.1</u>, must be done at the first follow-up visit after discontinuation at the latest.
- Research blood will be drawn at the time of disease progression.
- If a patient discontinues treatment without progressive disease and a new line of antineoplastic therapy is initiated, he/she will be censored for progression at that time point, research blood should be drawn, and AE/SAE follow up will cease.
- Upon disease progression or censoring for progression, the patient will be followed for survival per the progressive disease follow-up schedule in <u>Section 8.5.3</u>.

Follow-up will include collection of data of the following procedures. The procedures are not required every 8 weeks, but information from such procedures that are done per standard of care procedures will be collected if performed:

- Physical examination, including vital signs, weight and ECOG performance status
- Complete blood count, including platelets and differential
- Blood chemistries:
  - o BUN, creatinine, electrolytes (K+, Na+, Cl-, CO2), glucose, calcium, magnesium
- Liver function tests:
  - Total protein, albumin, total bilirubin, AST (SGOT), ALT (SGPT), and alkaline phosphatase

- Adverse event follow-up per <u>Section 8.5.1</u>.
- Survival Assessment
- Research blood for correlative studies at the time of disease progression as noted above.
- Tumor measurements according to RECIST 1.1

## 8.5.3 Progressive disease follow-up

Patients who discontinue treatment with progressive disease, experience progression during non-progressive disease follow up, or are censored for progression, will be followed for survival every 12 weeks (+/- 2 weeks) for 2 years.

AE/SAE assessment will be performed by phone contact or per a standard of care visit at least 60 days after the last dose of study drug, and per the requirements in <u>Section 8.5.1</u>.

#### 9. BIOMARKER, CORRELATIVE, OR SPECIAL STUDIES

Any remaining biospecimens collected for the research will be placed in a biorepository if subjects agree and consent to future use of their samples.

## 9.1 Submission of archived diagnostic tissue

For randomized subjects, submission of primary tumor tissue blocks (or slides, if blocks are not available) from procedures **prior to clinical cetuximab exposure** should be submitted for biomarker correlatives. This includes: A representative paraffin block of the original diagnosis and/or any repeat diagnostic biopsies, if available. Include a copy of the corresponding pathology report with the archived tissue. Collection, preparation, and shipping information for the archived tissue is in the Lab Manual. All efforts must be made to obtain paraffin blocks. If paraffin blocks are not available or the pathology department will only release slides, please contact the Sponsor-Investigator prior to requesting slides. A 3 mm core, punched from the tissue block with a punch tool, and 5-10 unstained slides of 5 micron thickness mounted on positively-charged glass slides may be acceptable.

#### 9.2 Research biopsy

All patients will be evaluated for a research biopsy at the time of enrollment. The biopsy is to be done prior to initiation of protocol treatment. Biopsies of primary tumor, accessible metastatic tumor, cutaneous lesion, or lymph node can occur in the outpatient office of the head and neck surgeon, with local anesthetic per standard of care. Biopsies of lymph nodes requiring imaging

guidance or distant metastases will occur under the care of an interventional radiologist, with ultrasound or CT guidance and local anesthetic per standard of care.

Omission of the research biopsy is allowed if performing the biopsy is not safe and/or feasible, and/or would present unacceptable clinical risk. Contact the Sponsor-Investigator for approval to omit the research biopsy. If the research biopsy is omitted, archived tumor tissue should be collected to substitute for the lack of baseline tissue. The archived tissue substituted for the Research Biopsy should be the **most recent** biopsy available and the corresponding pathology report must be obtained. (Substitution of archived tumor tissue for the research biopsy is independent of the archived tissue submission described above in <u>Section 9.1.)</u>

## 9.2.1 Research Biopsy Methodology

Research biopsies will consist of a cup forceps biopsy, a core needle biopsy, or a punch biopsy that can be safely performed in the outpatient setting with only local anesthesia. During the biopsy procedure, at least two cores of tissue 1-cm in length should be obtained with an 18-guage core biopsy needle (18-gauge or greater is preferred; 20-gauge is acceptable) – or the equivalent with cup forceps biopsy.

Collection, preparation, and shipping information for the research biopsy is in the Lab Manual.

#### 9.3 Research Blood

Blood for research purposes will be collected at the following time points:

- baseline
- end of cycles when a tumor assessment is due (Refer to Section 8.3.2 and Section 8.3.3)
- at the end of treatment if not collected within the prior 14 days
- at disease progression if not collected within the prior 14 days

Peripheral blood obtained by venipuncture will serve as the source for laboratory testing. Up to 70 mL of blood may be obtained at each draw. See the Lab Manual for collection information. Research blood will be used for correlative research and will be batch processed.

#### **10.STATISTICAL METHODS**

#### 10.1 Study Design

This is an open-label phase II trial with a randomized, non-comparative, two-arm design (Arm A: ficlatuzumab vs. Arm B: ficlatuzumab + cetuximab) in patients with recurrent and/or metastatic head and neck squamous cell carcinoma after failure of anti-EGFR therapy.

## **10.2** Primary Objective

The primary objective is to estimate the efficacy of ficlatuzumab, with or without cetuximab, as measured by the endpoint of PFS. Patients will be evaluable for PFS from the time of their first treatment with ficlatuzumab. PFS will be measured from the date of randomization until the date of progression or death. Patients without progression will be censored at the date of last follow up.

## **10.3** Sample Size Determination

The primary objective of this study is to estimate PFS in both arms. The sample size calculation thus is based on the primary endpoint of PFS. Given no data are available for single-agent ficlatuzumab in patients with recurrent and/or metastatic HNSCC refractory to platinum, cetuximab, and PD-1 inhibition, the historical control will be represented by dealer's choice chemotherapy in the phase III trial of nivolumab in platinum-refractory HNSCC: 2 months. This median PFS is very similar to single-agent data in the refractory, recurrent and/or metastatic setting for cetuximab, afatinib, and methotrexate <sup>49, 50</sup>. We would like to investigate whether the new regimen in either arm can improve the median PFS from 2 months to 3.33 months (i.e. 60% improvement in median PFS). To detect such an improvement, the study design requires 66 eligible patients (33 eligible patients on each arm) over 24 months with an additional follow-up of 6 months (making the study duration of approximately 2.5 years in total), using a log-rank test with 90% power while assuming a 0.10 one-sided type 1 error rate. Full information for the primary endpoint of PFS will occur at 33 events per arm. To account for an assumed 10% ineligibility/drop-out rate, 74 patients in total will be accrued to obtain the necessary 66 eligible randomized patients. If one arm achieves the hypothesized median PFS, that arm will be advanced to phase III testing. If both arms achieve the hypothesized PFS, the numerically superior arm will be advanced to phase III testing.

Definition of Evaluable:

Subjects who receive at least one dose of ficlatuzumab will be considered evaluable.

#### 10.4 Secondary Objectives

The secondary objectives of this trial are to describe toxicity and, to obtain additional measures of efficacy including response rate and overall survival.

#### **10.4.1 Toxicity**

Patients will be evaluable for toxicity from the time of their first treatment with ficlatuzumab. The proportion of AEs will be reported in accordance with NCI CTCAE v.4.0 grading criteria.

#### **10.4.2 Other Efficacy Endpoints**

Response rate will be assessed by modified RECIST criteria, version 1.1. Overall survival will be measured from the date of randomization until the date of death.

## 10.5 Exploratory Objectives

The exploratory objectives of this trial are to describe patient reported quality of life and to evaluate whether candidate biomarkers are prognostic in the context of treatment with ficialtyzumab.

## **10.5.1 Patient-Reported Outcomes**

Quality of life will be described according to FACT-H&N Symptom Index scores obtained at baseline and after two cycles of study treatment.

## **10.5.2 Biomarker endpoints**

We will evaluate the relationship between clinical outcomes (PFS, RR) and candidate tumoral, genomic, peripheral, and immune biomarkers, potentially including but not limited to: tumor HGF and cMet expression; mutations in *PIK3CA*, *PTEN*, and *HRAS*; peripheral serum biomarkers including HGF, soluble HGF, and IL6; peripheral lymphocyte populations; archived and baseline immune infiltrate.

Two candidate mechanistic biomarkers will be prioritized for specialized alpha spending: 1) baseline HGF expression; 2) baseline cMet expression. Testing two biomarkers each at  $\alpha = .05$  guarantees a maximum 10% false discovery rate for this exploratory objective.

Other candidate biomarkers in tumor and blood described above will be quantitatively measured and will be evaluated as predictors of PFS and/or tumor response in appropriate generalized linear models. Calculated p values for testing the significance of the prediction models will be adjusted for false discovery by the method of Benjamini and Hochberg.<sup>51</sup>

#### 10.6 Statistical Analysis Plan

Progression-free and overall survival will be estimated for each arm using a Kaplan-Meier curve. Toxicities and the response rate will be tabulated and reported with 95% exact confidence intervals. The relationship between progression-free survival and the candidate biomarkers will be assessed using Cox proportional hazards models. The relationship with clinical response will be assessed using logistic regression models.

## **10.7 Continuous Monitoring Rule for Futility**

The study will include a continuous Bayesian monitoring rule for futility. We will accrue and observe the first 8 evaluable patients on each arm, then continuously observe the proportion of patients who are without progression at 16-weeks. Based on the hypothesized increase in median progression-free survival from the historical rate of 2 months to 3.33 months in either the ficlatuzumab arm or the ficlatuzumab plus cetuximab arm, the expected proportion

progression-free at 16 weeks would be 0.46 under the alternative hypothesis. A Bayesian predictive probability design was used to estimate the rejection regions to stop an arm for futility.<sup>52</sup> The rejection regions to stop an arm for futility are: 0/8, 1/9, 2/13, 3/16, 4/19, 5/21, 6/24, 7/26, 8/28, 9/29, 10/31, 11/32, 12/33. Thus, if none of the first 8 patients is progression-free at 16 weeks, that arm will be stopped, or if only 1 of the first 9 patients is progression-free, that arm will be stopped, etc. This design has 80% power at  $\alpha = 0.10$  with an expected sample size of 21.3 under the null hypothesis and 31.4 under the alternative hypothesis. The probability of early termination under the null hypothesis is 0.86. The rejection regions were derived to maximize power under the alternative hypothesis. There was no Bayesian predictive probability design with 90% statistical power given the proposed median survival times and sample size with  $\alpha = 0.10$ .

#### 11. DATA SAFETY MONITORING PLAN

## 11.1 Identification of the DSMB obligated for oversight responsibilities

Dr. Julie Bauman at the University of Arizona Cancer Center (UACC) will assume the role of the Sponsor. The UACC Data and Safety Monitoring Board (DSMB) will assume responsibility for oversight of safety monitoring. Based on the UACC DSMB Charter this is a high risk study.

## 11.2 Identification of the entity obligated and requirements for routine monitoring duties

Affiliate sites that participate in this trial will choose, through a reciprocal agreement with UACC, either to:

- 1) Perform monitoring per the sites' Data and Safety Monitoring Plan, only if the site has fully approved NCI Data and Safety Monitoring Plan.
- 2) Allow UACC to conduct remote and on-site monitoring for this trial in accordance with the UACC's approved NCI Data and Safety Monitoring Charter/Monitoring Plan.
- 3) Perform monitoring per the UACC's Data and Safety Monitoring Charter/Plan.

If a site-specific monitoring plan will be used, the UACC DSMB must review the sites' Data and Safety Monitoring Plan and approve that the plan is acceptable. If the UACC DSMB finds that a plan is not acceptable, the UACC or the site's internal monitors will perform monitoring per the UACC Data and Safety Monitoring Plan.

Elements that are required to be included within each site-specific DSM plan are:

- A process to verify eligibility by the local monitoring team.
- Frequency and extent of monitoring activities for this trial at the site

#### 11.3 Monitoring progress, assuring data accuracy and protocol compliance

Frequency and methodology of routine monitoring may vary slightly from institution to institution.

Regardless of monitoring entity, all monitoring reports must be completed and submitted to the local site PI, the Sponsor-Investigator, and UACC DSMB.

All submitted serious adverse events will be submitted to the UACC DSMB Coordinator monthly and then reviewed by the DSMB Chair.

Any identified SAE trends will be made available for review at the investigator teleconferences.

A teleconference will occur on a regular schedule to review study progress and any safety, or other, issues. Minutes of these teleconference meetings will be submitted to UACC DSMB for review.

At each site, the Principal Investigator will ensure the accuracy, completeness, legibility and timeliness of the data reported in the OnCore electronic Case Report Form (eCRF), and other data formats. Source documentation supporting the study data should indicate the subject's participation in the trial and should document the dates and details of study procedures, adverse events, and patient status.

Case report forms, which include adverse event forms, serious adverse event forms, and protocol or patient deviations must be completed via the UACC OnCore CRM database.

#### 11.4 Oversight Activities by the UACC DSMB

Any identified safety issue will be submitted to the UA IRB, DSMB or other oversight entity as applicable. In addition to review of site specific monitoring, the convened UACC DSMB will review all monitoring reports and findings every 6 months. Every 6 months, the UACC convened DSMB will perform a review of all study data which will include the following:

- SAEs
- AEs
- Protocol Deviations
- Any pending action items (i.e., responses to DSMB reports; pending items from routine monitoring reports).

Study activity and safety information will be routinely submitted to the UACC DSMB.

In addition to site specific monitoring, the local PI will complete a status report for each UACC DSMB review. These reports should include summaries of:

- Study activity, cumulative and for the period under review;
- Safety information (non-serious and serious adverse events);
- Status of study in relationship to stopping rules;
- Routine monitoring and protocol compliance (describe the monitoring process and identify the status of the monitoring);
- Attachments (AE data reviewed by the PI to compile the report, SAE reports, results of any review(s), applicable correspondence with the IRB or other regulatory agencies.

Data and Safety Monitoring Board determinations will be reported to the University of Arizona IRB at least annually. DSMB determinations will be distributed to the sites contemporaneously.

## 11.5 Process to implement study closure when significant risks or benefits are identified

This study may be prematurely terminated, if in the opinion of the investigator or Aveo, there is sufficient reasonable cause. Written notification documenting the reason for study termination will be provided to the investigator or Aveo by the terminating party.

Circumstances that may warrant termination include, but are not limited to:

- Determination of unexpected, significant, or unacceptable risk to patients
- Failure to enter patients at an acceptable rate
- Insufficient adherence to protocol requirements
- Insufficient complete and/or evaluable data
- Plans to modify, suspend or discontinue the development of the drug

Should the study be closed prematurely, remaining study drug must be returned to Aveo or destroyed.

#### 11.6 Identification of the sponsor or funding agency, as applicable

Dr. Julie E. Bauman is the sponsor-investigator responsible for all requirements as set out in 21 CFR 312. Aveo Oncology provides support for the trial by providing the investigational product.

 v10, 05/23/2023

The sponsor-investigator will immediately notify applicable entities of any action resulting in a temporary or permanent suspension of the study.

#### 12.ADVERSE EVENT REPORTING

#### 12.1 Definitions

The following definitions of terms apply to this section:

<u>Adverse event</u>: Any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. The term "Adverse Event" is inclusive of SAEs.

<u>Life-threatening adverse event or life-threatening suspected adverse reaction</u>: An adverse event or suspected adverse reaction is considered "life-threatening" if, in the view of either the investigator or sponsor, its occurrence places the patient or subject at immediate risk of death. It does not include an adverse event or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.

<u>Serious adverse event</u>: An adverse event is considered "serious" if it results in any of the following outcomes:

- death,
- a life-threatening adverse event,
- inpatient hospitalization or prolongation of existing hospitalization,
- a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or
- a congenital anomaly/birth defect.
- Important medical events that may not result in death, be life-threatening, or require
  hospitalization may be considered serious when, based upon appropriate medical
  judgment, they may jeopardize the patient or subject and may require medical or
  surgical intervention to prevent one of the outcomes listed in this definition.
- Pregnancy

<u>Suspected adverse reaction</u>: Any adverse event for which there is a reasonable possibility that the drug caused the adverse event. For the purposes of IND safety reporting, "reasonable possibility" means there is evidence to suggest a causal relationship between the drug and the adverse event. Suspected adverse reaction implies a lesser degree of certainty about causality than adverse reaction, which means any adverse event caused by a drug.

<u>Unexpected adverse event or unexpected suspected adverse reaction</u>: An adverse event or suspected adverse reaction is considered "unexpected" if it is not listed in the investigator brochure or is not listed at the specificity or severity that has been observed; or, if an

investigator brochure is not required or available, is not consistent with the risk information described in the general investigational plan or elsewhere in the current application, as amended. For example, under this definition, hepatic necrosis would be unexpected (by virtue of greater severity) if the investigator brochure referred only to elevated hepatic enzymes or hepatitis. Similarly, cerebral thromboembolism and cerebral vasculitis would be unexpected (by virtue of greater specificity) if the investigator brochure listed only cerebral vascular accidents. "Unexpected," as used in this definition, also refers to adverse events or suspected adverse reactions that are mentioned in the investigator brochure as occurring with a class of drugs or as anticipated from the pharmacological properties of the drug, but are not specifically mentioned as occurring with the particular drug under investigation.

## 12.2 Description of Adverse Event Reporting Procedures

Adverse events will be recorded in the adverse events record form in the UACC OnCore CRM and reviewed by the local Principal Investigator. All Adverse Events as defined in this section will be collected starting on Cycle 1, Day 1 must be recorded. AEs will be followed per the details indicated in protocol <u>Section 8.5.1</u>. Only AEs meeting one of the following criteria will be entered into the OnCore CRM study database:

- Any AE that is Grade 3 or higher, regardless of relationship to the study drug
- Any AE that results in submission of a Serious Adverse Event (i.e., hospitalization for a non-serious grade AE)
- Any intolerable (per the opinion of the treating investigator) Grade 2 AE
- Any Grade AE resulting in a dose reduction of ficlatuzumab or cetuximab
- Any Grade 2 laboratory or vital sign values that are deemed clinically significant by the treating investigator
- Any Grade AE in the following categories of interest:
  - o Rash
  - Diarrhea
  - o Edema, peripheral
  - o Edema, head, face and neck
  - o Hypoalbuminemia

All adverse events will be classified using either the MedDRA term or NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 and will address:

- Grade
- Relationship to ficiatuzumab (not related, unlikely, possible, probable, definitely)
- Relationship to cetuximab (not related, unlikely, possible, probable, definitely)

- Causality other than study drug (disease related, concomitant medication related, intercurrent illness, other)
- Date of onset
- Date of resolution
- Frequency of event (single, intermittent, continuous)
- Event outcome (resolved, ongoing, death)
- Action taken with ficlatuzumab (none, held, dose reduced, discontinued, medication given)
- Action taken with cetuximab (none, held, dose reduced, discontinued, medication given)

## 12.3 Reporting of Serious Adverse Events

All Serious Adverse Events as defined in <u>Section 12.1</u> will be collected starting Cycle 1, Day 1 and must be reported to the Sponsor. SAEs will be followed per the details indicated in protocol <u>Section 8.5.1</u>. SAEs must be reported to the IRB of Record per local procedure.

Regardless of attribution, SAEs must be reported to the sponsor and the UACC DSMB within 24 hours of notification of the event. SAEs will also be copied to the Aveo pharmacovigilance entity, Parexel. The FiclaYCetux Serious Adverse Event Report Form must be used to report SAEs and redacted, relevant medical records must be attached when available. Follow-up information that describes an increase in severity or risk must be submitted within 24 hours of notification of the information. Follow-up SAE reports must also be reported within 24 hours of notification of updated information related to the event.

The Sponsor, UACC DSMB, and/or the Aveo pharmacovigilance entity, Parexel, may contact site personnel with queries to ensure all necessary information is obtained.

SAEs must be recorded in the OnCore "SAEs" tab.

#### 12.4 Review of Safety Information: Sponsor-Investigator Responsibilities

The sponsor will review all SAEs and safety information received to determine if the events meet the reporting requirements for FDA. Information will be reviewed and reported, if needed, by the Sponsor-Investigator consistent with 21 CFR 312.32 IND safety reporting.

## 12.5 IND safety reports for ficlatuzumab

Suspected, Unexpected, and Serious Adverse Drug Reaction (SUSAR)/IND Safety reports received from Aveo will be distributed to site investigators within 15 days of receipt. Any updates to the ficial fiction and Investigator Brochure will be distributed upon receipt from Aveo.

#### 13. DATA HANDLING AND RECORD-KEEPING

Local site PIs are responsible to maintain, archive, and retain research records according to local and Federal policy, and per the Clinical Trial Agreement. This includes, but is not limited to, accurate drug accountability and disposition records, case histories, and source documents.

The Sponsor-Investigator will maintain records in accordance with Good Clinical Practice guidelines.

The Sponsor-Investigator will retain the specified records and reports for up to 2 years after the marketing application is approved for the investigational drug; or, if a marketing application is not submitted or approved for the investigational drug, until 2 years after investigations under the IND have been discontinued and the FDA so notified.

#### 14.ETHICS AND REGULATORY COMPLIANCE

## 14.1 Institutional Review Board (IRB) approval

The Sponsor-Investigator will obtain, from the University of Arizona (UA) Institutional Review Board (IRB), prospective approval of the clinical protocol and corresponding informed consent form(s); modifications to the clinical protocol and corresponding informed consent forms, and advertisements (i.e., directed at potential research subjects) for study recruitment. Once UA IRB approval is secured, the revised materials will be distributed to each participating site. Each site participating in the trial must obtain IRB approval from the applicable IRB prior to initiating the research.

The only circumstance in which a deviation from the current IRB-approved clinical protocol/consent form(s) may be initiated in the absence of prospective IRB approval is to eliminate an apparent immediate hazard to the research subject(s). Per local procedure, investigators must promptly notify the applicable IRB of the deviation.

The University of Arizona IRB operates in compliance with FDA regulations at <u>21 CFR Parts 50</u> and <u>21 CFR 56</u>, and in conformance with applicable International Conference on Harmonization (ICH) Guidelines on Good Clinical Practice (CGP).

In the event that the University of Arizona IRB requires, as a condition of approval, substantial changes to a clinical protocol submitted under an FDA-accepted IND application, or in the event of the Sponsor-Investigator's decision to modify the previously accepted clinical protocol:

• The Sponsor-Investigator will submit (i.e., in advance of implementing the change) a Protocol Amendment to the IND describing any change to a Phase 2 or Phase 3 protocol that significantly affects the safety of subjects, the scope of the investigation, or the

scientific quality of the study. Examples of Phase 2 and 3 clinical protocol changes requiring the submission of a Protocol Amendment include:

- o Any increase in drug dosage or duration of exposure of individual subjects to the investigational drug beyond that described in the current protocol, or any significant increase in the number of subjects under study.
- o Any significant change in the design of the protocol (such as the addition or deletion of a control group).
- o The addition of a new test or procedure that is intended to improve monitoring for, or reduce the risk of, a side effect or adverse event; or the dropping of a test intended to monitor the safety of the investigational drug.

## 14.2 Ethical and scientific conduct of the clinical research study

The clinical research study will be conducted in accordance with the current IRB-approved clinical protocol; ICH GCP Guidelines adopted by the FDA; and relevant policies, requirements, and regulations of the University of Arizona IRB and applicable federal agencies.

## 14.3 Subject informed consent

The Sponsor-Investigator and local site PIs will make certain that an appropriate informed consent process is in place to ensure that potential research subjects, or their authorized representatives, are fully informed about the nature and objectives of the clinical study, the potential risks and benefits of study participation, and their rights as research subjects. The site PIs or a sub-investigator(s) designated appropriately, will obtain the written, signed informed consent of each subject, or the subject's authorized representative, prior to performing any study-specific procedures on the subject. The date and time that the subject, or the subject's authorized representative, signs the informed consent form and a narrative of the issues discussed during the informed consent process will be documented in the subject's case history. Each site will retain the original copy of the signed informed consent form, and a copy will be provided to the subject, or to the subject's authorized representative.

The site Pls/sub-investigators will make certain that appropriate processes and procedures are in place to ensure that ongoing questions and concerns of enrolled subjects are adequately addressed and that the subjects are informed of any new information that may affect their decision to continue participation in the clinical study. In the event of substantial changes to the clinical study or the risk-to-benefit ratio of study participation, a revised informed consent will be presented to each enroll subjects for their consideration regarding continued participation in the clinical study. A subject can withdraw from the study at any time.

## 14.4 Confidentiality

All records identifying subjects must be kept confidential per local and Federal policy. Minimum necessary standards must be followed. Information sent to the Sponsor must be redacted. Site Pls must maintain a list of subjects and assigned study ID numbers to enable identification of the patients. Subject identities will not be used in any results that are published.



## FiclaYCetux Protocol Signature Page Protocol Version: 8

## **Investigator Agreement**

STUDY TITLE: A Randomized, Phase II Study of Ficlatuzumab with or without Cetuximab in Patients with Cetuximab-Resistant, Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma

By signing below I agree:

- 1) That my staff and I have read, understand and will adhere to the protocol as written, and that any changes to the protocol will be agreed to and approved by the Principal Investigator and the Institutional Review Board (IRB)
- 2) To abide by all obligations stated on the FDA Form 1572 and other documents required by regulation;
- 3) To conduct this study in accordance with the current International Conference on Harmonization (ICH) guidance, the Good Clinical Practices (GCP) guidance, the Declaration of Helsinki, US FDA regulations and local IRB and legal requirements;
- 4) To obtain IRB approval of the protocol, any amendments to the protocol, and periodic reapproval as required, and to keep the IRB informed of adverse events as required by their guidelines report the status of the study to them;
- 5) To ensure that each individual enrolled into the trial, or legally authorized representative, has read, understands, and has signed the Informed Consent form;
- 6) To ensure that I and all persons assisting me with the study are adequately informed and trained about the study and the possible adverse events associated with the study required medication
- 7) To make prompt reports of SAEs and deaths to the Sponsor/FDA according to the regulations;
- 8) To prepare and maintain adequate and accurate case histories to document all observations and other data pertinent to the study for each individual enrolled in the clinical trial.

| Site Principal Investigator Signature | Date |
|---------------------------------------|------|
| Investigator Name (Print) | |

#### 15.APPENDICES

## 15.1 Appendix A: FACT-H&N Symptom index (FHNSI)

| Subject ID: | Subject Initials: | Date Completed: |
|-------------|-------------------|-----------------|
|-------------|-------------------|-----------------|

#### FACT/NCCN HNSI

Below is a list of statements that other people with your illness have said are important. Please circle or mark one number per line to indicate your response as it applies to the <u>past 7 days</u>.

| | l | Not at<br>all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|
| GP4 | I have pain | 0 | 1 | 2 | 3 | 4 |
| GP1 | I have a lack of energy | 0 | 1 | 2 | 3 | 4 |
| HAN7 | I can swallow naturally and easily | 0 | 1 | 2 | 3 | 4 |
| HAN 12 | I have pain in my mouth, throat or neck | 0 | 1 | 2 | 3 | 4 |
| HAN3 | I have trouble breathing | 0 | 1 | 2 | 3 | 4 |
| HAN10 | I am able to communicate with others | 0 | 1 | 2 | 3 | 4 |
| GP2 | I have nausea | 0 | 1 | 2 | 3 | 4 |
| HAN11 | I can eat solid foods | 0 | 1 | 2 | 3 | 4 |
| GES | I worry that my condition will get worse | 0 | 1 | 2 | 3 | 4 |
| GF7 | I am content with the quality of my life right now | 0 | 1 | 2 | 3 | 4 |

| English (Universal)<br>Version 4, Copyright 2001 | | | 22 Ay<br>Page | pril 2020<br>e 1 of 1 |
|---|---|---|---|---|
| For Internal Use ONLY | | | | |
| Form Completed By: | Subject | Other (name): | Sign/Date: | |
| Comment, if applicable: | | | | |

## 15.2 Appendix B: Performance Status Criteria

| ECC | OG Performance Status Scale | Karr | nofsky Performance Scale |
|---|---|---|---|
| Grade | Descriptions | Percent | Description |
| | Normal activity. Fully active, able | 100 | Normal, no complaints, no evidence of disease. |
| 0 | to carry on all pre-disease performance without restriction. | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| 1 | Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able | 80 | Normal activity with effort; some signs or symptoms of disease. |
| I | to carry out work of a light or sedentary nature ( <i>e.g.</i> , light housework, office work). | 70 | Cares for self, unable to carry on normal activity or to do active work. |
| 2 | In bed <50% of the time. Ambulatory and capable of all | 60 | Requires occasional assistance, but is able to care for most of his/her needs. |
| 2 | self-care, but unable to carry out<br>any work activities. Up and about<br>more than 50% of waking hours. | 50 | Requires considerable assistance and frequent medical care. |
| | In bed >50% of the time. | 40 | Disabled, requires special care and assistance. |
| 3 | Capable of only limited self-care, confined to bed or chair more than 50% of waking hours. | 30 | Severely disabled,<br>hospitalization indicated. Death<br>not imminent. |
| 4 | 100% bedridden. Completely disabled. Cannot carry on any | 20 | Very sick, hospitalization indicated. Death not imminent. |
| 4 | self-care. Totally confined to bed or chair. | 10 | Moribund, fatal processes progressing rapidly. |
| 5 | Dead. | 0 | Dead. |

15.3 Appendix C: Study Calendar (Also see Section 8)

| | Screening | - | Study Treatme | ent | | Falls | ما ا س |
|---|---|---|---|---|---|---|---|
| | Within 28 | | 28 Day Cycles | ; 2 | | FOIIC | оw Up |
| | days of<br>registration<br>(except<br>pregnancy<br>within 14 days<br>of registration) | Day 1<br>+/- 3 days | Day 15<br>+/- 3 days | Every 8<br>weeks <sup>13</sup><br>Day 28<br>+/- 7 days<br>(C12+ Optional<br>q12wks +/- 14d) | End Of<br>Treatment <sup>1</sup> | Non-PD<br>Follow-<br>up <sup>3</sup><br>q8wks<br>+/- 2<br>week | PD<br>Follow-<br>up <sup>19</sup><br>q12wks<br>+/- 2<br>weeks |
| Medical History | Х | | | | | | |
| Physical Exam & Vital Signs | Х | Х | Х | | Х | Z | |
| Height | Х | | | | | | |
| Weight | Х | X <sup>4</sup> | X <sup>4</sup> | | Х | Z | |
| ECOG Performance Status | Х | Х | Х | | Х | Z | |
| CBC with Differential <sup>5</sup> | Х | Х | Х | | Х | Z | |
| Serum chemistries and Liver function tests <sup>5</sup> | Х | Х | Х | | Х | Z | |
| Magnesium <sup>5</sup> | X | Х | Х | | Х | Z | |
| Documentation of Corrected Calcium | Х | | | | | | |
| Research (correlatives) blood | X 6 | | | X <sup>7</sup> | X | X 8 | |
| Pregnancy test | X 9 | | | | | | |
| Research biopsy <sup>10</sup> | Х | | | | | | |
| Confirmation of availability of archived diagnostic specimens | X 11 | | | | | | |
| Tumor measurements,<br>RECIST 1.1 (CT or MRI) <sup>12</sup> | Х | | | X <sup>13</sup> | X | Z | |
| FACT-H&N Symptom Index | X 6 | | | X <sup>14</sup> | X 14 | | |
| Tobacco Assessment | X 6 | | | | | | |
| Oropharyngeal & unknown primary cases, p16 Status 15 | Х | | | | | | |
| Registration/Randomization | Х | | | | | | |
| Cetuximab | | Х | Х | | | | |
| Ficlatuzumab | | X | Х | | | | |
| Concomitant medication review | Х | Х | Х | | Х | | |
| Adverse event evaluation | | Х | Х | | X <sup>16</sup> | X <sup>17</sup> | X 18 |
| Survival assessment | | | | | | Х | X <sup>19</sup> |

 v10, 05/23/2023

- <sup>5</sup> May be performed on the day of, or within the 3 days prior to study treatment.
- <sup>6</sup> May be performed during screening, or prior to drug administration on Cycle 1, Day 1.
- <sup>7</sup> For convenience, research blood may be drawn simultaneously with pre-treatment labs for the next cycle. *Subjects who transition to every-12-week tumor assessments will have the research blood drawn every 12 weeks, consistent with the tumor assessment schedule. Refer to Section 8.3.3*
- <sup>8</sup> Research blood will be obtained at the time of disease progression or censored for progression (see footnote 3 above, and <u>Section 8.5.2</u>) during the follow up period, then followed per the progressive disease follow up.
- <sup>9</sup> A negative pregnancy test is required in women of child-bearing potential within 14 days prior to registration. Negative pregnancy test must be confirmed again within 3 days prior to first drug administration.
- <sup>10</sup> Archived tumor tissue, preferably the most recent tissue available, may be substituted if the biopsy is not safe and/or feasible, and/or would present unacceptable clinical risk, and the Sponsor has approved omission of the baseline biopsy. See <u>Section 9.2</u>.
- <sup>11</sup> Archived tissue, preferably primary tumor tissue blocks (or slides, if blocks are not available) from procedures **prior to clinical cetuximab exposure.** This is not an eligibility requirement and subjects can be randomized without this confirmation.
- <sup>12</sup> For scheduling convenience, tumor measurements may occur on day 1 of the following cycle, so long as the scan is done and results are known **prior** to drug administration.
- <sup>13</sup> Tumor measurements must be performed every 8 weeks, +/- 7 days, regardless of any delay that occurs within the prior 2 cycles. Subjects who remain on treatment past Cycle 12 can transition to tumor assessments being performed every 12 weeks, +/- 14 days. Refer to <u>Section 8.3.3</u>.
- <sup>14</sup> FACT-H&N Symptom Index will be performed at baseline and at the end of cycle 2 and cycle 6 only, or when the subject is censored for progression after C4D28 but before C6D28 (see <u>EOT procedures</u>). For scheduling convenience, FACT-H&N Symptom Index may be completed on day 1 of the following cycle or at the EOT visit.
- <sup>15</sup> For oropharyngeal & unknown primary, p16 status must be established, if not previously known, before randomization.
- <sup>16</sup> Subject will be followed for AEs/SAEs for 60 days **after last dose of study drug** or until the initiation of subsequent antineoplastic therapy, whichever is earlier. (Refer to protocol <u>Section 8.5.1</u> for important and specific details on collection and follow up of AEs.)
- <sup>17</sup> Subjects who end treatment **due to a reason other than progressive disease** will have an AE assessment at the first follow-up visit. (Refer to protocol <u>Section 8.5.1</u> for important and specific details on collection and follow up of AEs.)
- <sup>18</sup> Subjects who end treatment **due to progressive disease** will have an AE assessment at least 60 days after last dose of study drug. (Refer to protocol <u>Section 8.5.1</u> for important and specific details on collection and follow up of AEs.)
- <sup>19</sup> Subjects will be followed for survival for 2 years after disease progression.

<sup>&</sup>lt;sup>1</sup> The End of Treatment visit should be performed as soon as possible, but preferably within 30 days after the off-treatment decision date. Procedures will be performed if not performed in the previous 14 days, except tumor measurements should only be performed if not performed in the previous 28 days and only if it is an appropriate standard of care procedure.

<sup>&</sup>lt;sup>2</sup> Refer to <u>Section 5.5.1</u> which addresses scheduling when there are missed and/or skipped visits due to treatment delays or other.

<sup>&</sup>lt;sup>3</sup> Procedures indicated with "Z" are not required to be performed for the research, but if they are performed for standard of care, the data will be collected. Patients who initiate a new line of antineoplastic therapy will be censored for progression at that time point; research blood will be drawn and they will be followed per the progressive disease follow-up schedule.

<sup>&</sup>lt;sup>4</sup> For both agents: Recalculate the doses of both ficiatuzumab and cetuximab only if there is a ≥ 10% change in weight. Exception: If, in the opinion of the treating investigator, weight change of ≥ 10% is due to edema, recalculation of the ficiatuzumab dose is not required. This decision must be clearly documented. Refer to Section 5.

## 15.4 Appendix D: Tobacco Use Assessment Form

| | | Resistant, Rect | urrent/Metastatic Head an | d Neck Squamous | Cell Carcinoma | |
|---|---|---|---|---|---|---|
| | | | Tobacco Use Asse | ssment Form | | |
| 1. | Have you | ever smoked a | total of 100 eigarettes (ap | proximately 5 pac | cks) or more over your l | ife-time |
| | ☐ Ye | s 🗌 No | | | | |
| | If no, ski | p to question 6 | 5. | | | |
| 2. | Have you<br>longer? | ever smoked c | rigarettes regularly, that is, | at least one cigar | ette per day for six mon | ths or |
| | ☐ Ye | s 🗌 No | | | | |
| 3 | | | you first started smoking | at least one cinare | ette ner dav? | |
| | | ears old | , you make a smoking | an reast one eigare | nto per day: | |
| 4 | | arrently smoke | cigarettes" | | | |
| | ☐ Ye | s 🗆 No | | | | |
| | If | no, how old we | ere you when you <u>last</u> smo | ked a cigarette? | | |
| | | years old | | | | |
| 5. | | | ears that you have smoked | , how many cigare | ettes do you (or did you) | usually |
| | smoke in | | | | | |
| | | o 9 cigarettes pe<br>to 19 cigarettes | | | | |
| | 20 | to 29 cigarettes<br>to 39 cigarettes | s per day | | | |
| | | to 49 cigarettes | | | | |
| 6. | Have you | ever smoked e | rigars regularly, that is, at | least one cigar per | day for six months or le | mger? |
| | ☐ Ye | s 🗌 No | | | | |
| | If no, ski | p to question 1 | 10. | | | |
| 7. | How old | were you when | you first started smoking | at least one eigar | per day? | |
| | ye | ars old | | | | |
| Version 0 | Us: Assessm:<br>04/20/2020<br>Law Subj | | Subject Initials: | | | Page I of |
| Version 0 | 04/20/2020<br>Lago Subj | ect ID: | | r | | Page 1 of |
| Version 0 | tare Subj | ect ID: | | r | | Page I of |
| Version 0 | Do you ci | eet ID: | cigars? | | | Page I of |
| Version 0 | Do you ci | ect ID: | | | | Page I of |
| Version 0 | tuw Subjutuw Subjutu | ect ID: urrently smoke s | cigars?<br>ere you when you <u>last</u> smo | sked a cigar? | | Page I of |
| Version 0 | Lue Subj | eet ID: arrently smoke s | cigars? | sked a cigar? | | Page I of |
| Version 0 Floka Cet 8. | Do you co | ect ID: arrently smoke s | cigars?<br>ere you when you <u>last</u> smo<br>uu usually smoke in a day? | oked a cigar? | Onte Completed: | |
| Version 0 Floka Cet 8. | Do you co | eet ID: urrently smoke s | cigars?<br>ere you when you <u>last</u> smo | oked a cigar? | Onte Completed: | |
| Version 0 Floka Cet 8. | Do you ce If How man cig Have you | eet ID: urrently smoke s | cigars? ere you when you last sme the usually smoke in a day? a pipe regularly, that is, at | oked a cigar? | Onte Completed: | |
| Version 0 Field Cet 8. | Do you co | eet ID: arrently smoke No no, how old we years old ye eigars did you tars per day ever smoked a no questionnaire | cigars? ere you when you last sme the usually smoke in a day? a pipe regularly, that is, at | sked a cigar? | Onte Completed: | |
| Version 0 Field Cet 8. | Do you ce Ye If How man cig Have you Ye If no, the | eet ID: arrently smoke No no, how old we years old ye eigars did you tars per day ever smoked a no questionnaire | cigars? ere you when you last smo to usually smoke to a day? To pipe regularly, that is, at to is complete. | sked a cigar? | Onte Completed: | |
| Version to | Do you ce If How man cig Have you Ye If no, the | eet ID: | cigars? ere you when you last smo to usually smoke in a day? to pipe regularly, that is, at to is complete. you first started smoking | sked a cigar? | Onte Completed: | |
| Version to | Do you ce If How man cig Have you Ye If no, the | eet ID: urrently smoke s | cigars? ere you when you last smo to usually smoke in a day? to pipe regularly, that is, at to is complete. you first started smoking | sked a cigar? | Onte Completed: | |
| Version to | Do you ce If no, the How land Yes If no, the Do you ce Yes If no, the Yes Do you ce | eet ID: | cigars? ere you when you last smo to usually smoke in a day? to pipe regularly, that is, at to is complete. you first started smoking | sked a cigar?<br>least one pipe per<br>at least one pipe p | Onte Completed: | |
| Version to | Do you ce If no, the How land Yes If no, the Do you ce Yes If no, the Yes Do you ce | eet ID: | cigars? ere you when you last sme to usually smoke in a day? pipe regularly, that is, at is complete. you first started smoking a pipe? | sked a cigar?<br>least one pipe per<br>at least one pipe p | Onte Completed: | |
| Version 0 | Do you cu Ye If How man Gig Have you Ye to U Ye Find the to Ye Ye Thin, the How old Ye Ye Thin, the Thinking | ect ID: urrently smoke No no, how old we years old ye egars did you tars per day ever smoked a no questionnaire were you when ars old arrently smoke No no, how old we years old about all the ye | cigars? ere you when you last sme to usually smoke in a day? pipe regularly, that is, at is complete. you first started smoking a pipe? | eked a cigar? least one pipe per at least one pipe p | day for six months or le | nger? |
| Version 0 | Do you cu Ye If How man cig Have you Ye to U Ten, the To Do you cu Ye If Thinking, smoke in | ect ID: urrently smoke s | cigars? ere you when you last sme to usually smoke m a day? t pipe regularly, that is, at t is complete. tyou first started smoking a pipe? ere you when you last sme | eked a cigar? least one pipe per at least one pipe p | day for six months or le | nger? |
| Version 0 | Do you cu Ye If How man cig Have you Ye to U Ten, the To Do you cu Ye If Thinking, smoke in | ect ID: urrently smoke No no, how old we years old ye egars did you tars per day ever smoked a no questionnaire were you when ars old arrently smoke No no, how old we years old about all the ye | cigars? ere you when you last sme to usually smoke m a day? t pipe regularly, that is, at t is complete. tyou first started smoking a pipe? ere you when you last sme | eked a cigar? least one pipe per at least one pipe p | day for six months or le | nger? |
| Version 0 8. 9. 10 11 12 | Do you cu Co Subjet How manature in the How old year If How old year If How in the How in the How | eet ID: arrently smoke No no. how old we years old years old years old years per day ever smoked a no questionnaire were you when arrently smoke No years old about all the ye a day? | cigars? ere you when you last sme to usually smoke m a day? t pipe regularly, that is, at t is complete. tyou first started smoking a pipe? ere you when you last sme | eked a cigar? least one pipe per at least one pipe p | day for six months or le | nger? |
| Version 0 Version 0 8 9 10 11 12 | Do you ce Thou Manager How man How man How pour Ve If no, the how old yee Yee If no, the how old yee Thou how o | eet ID: arrently smoke No no. how old we years old years old years old years per day ever smoked a no questionnaire were you when arrently smoke No years old about all the ye a day? | cigars? ere you when you last sme to usually smoke in a day? pipe regularly, that is, at is complete, you first started smoking a pipe? ere you when you last sme ears that you have smoked | eked a cigar? least one pipe per at least one pipe p | day for six months or le | nger? |
| Version 0 Version 0 8 9 10 11 12 For 1 | Do you co | ect ID: | cigars? ere you when you last sme to usually smoke in a day? pipe regularly, that is, at is complete, you first started smoking a pipe? ere you when you last sme ears that you have smoked | eked a cigar? least one pipe per at least one pipe p | day for six months or lo | nger? |
| Version 0 8 9 10 11 12 For 1 Com | Do you co Ye How man cig ye Have you Ye If no, the do ye If f Thinking, smoke in pi | ect ID: | cigars? ere you when you last sme to usually smoke in a day? pipe regularly, that is, at is complete, you first started smoking a pipe? ere you when you last sme ears that you have smoked | eked a cigar? least one pipe per at least one pipe p | day for six months or lo | nger? |
| Version 0 8 9 10 11 12 For 1 Com | Do you cu Sabju Sa | ect ID: | cigars? ere you when you last sme to usually smoke in a day? pipe regularly, that is, at is complete, you first started smoking a pipe? ere you when you last sme ears that you have smoked | eked a cigar? least one pipe per at least one pipe p | day for six months or lo | |

#### 16. REFERENCES

- 1. Kamangar F, Dores GM, Anderson WF. Patterns of Cancer Incidence, Mortality, and Prevalence Across Five Continents: Defining Priorities to Reduce Cancer Disparities in Different Geographic Regions of the World. Journal of Clinical Oncology. 2006;24: 2137-2150.
- 2. Jemal A, Siegel R, Xu J, Ward E. Cancer statistics, 2010. CA Cancer J Clin. 2010;60: 277-300.
- 3. Hong WK, Schaefer S, Issell B, et al. A prospective randomized trial of methotrexate versus cisplatin in the treatment of recurrent squamous cell carcinoma of the head and neck. Cancer. 1983;52: 206-210.
- 4. Forastiere AA, Metch B, Schuller DE, et al. Randomized comparison of cisplatin plus fluorouracil and carboplatin plus fluorouracil versus methotrexate in advanced squamous-cell carcinoma of the head and neck: a Southwest Oncology Group study. J Clin Oncol. 1992;10: 1245-1251.
- 5. Rubin Grandis J, Melhem MF, Gooding WE, et al. Levels of TGF-alpha and EGFR protein in head and neck squamous cell carcinoma and patient survival. J Natl Cancer Inst. 1998;90: 824-832.
- 6. Chung CH, Ely K, McGavran L, et al. Increased epidermal growth factor receptor gene copy number is associated with poor prognosis in head and neck squamous cell carcinomas. J Clin Oncol. 2006;24: 4170-4176.
- 7. Vermorken JB, Mesia R, Rivera F, et al. Platinum-based chemotherapy plus cetuximab in head and neck cancer. N Engl J Med. 2008;359: 1116-1127.
- 8. Seiwert TY, Burtness B, Mehra R, et al. Safety and clinical activity of pembrolizumab for treatment of recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-012): an open-label, multicentre, phase 1b trial. Lancet Oncol. 2016;17: 956-965.
- 9. Ferris RL, Blumenschein GR, Fayette J, et al. Further evaluations of nivolumab versus investigator's choice chemotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck: CheckMate 141. J Clin Oncol. 2016;34.
- 10. Ciardiello F, Tortora G. Epidermal growth factor receptor (EGFR) as a target in cancer therapy: understanding the role of receptor expression and other molecular determinants that could influence the response to anti-EGFR drugs. European Journal of Cancer. 2003;39: 1348-1354.
- 11. Grandis JR, Melhem MF, Barnes EL, Tweardy DJ. Quantitative immunohistochemical analysis of transforming growth factor- $\alpha$  and epidermal growth factor receptor in patients with squamous cell carcinoma of the head and neck. Cancer. 1996;78: 1284-1292.
- 12. Dassonville O, Formento JL, Francoual M, et al. Expression of epidermal growth factor receptor and survival in upper aerodigestive tract cancer. Journal of Clinical Oncology. 1993;11: 1873-1878.
- 13. Chung CH, Zhang Q, Hammond EM, et al. Integrating epidermal growth factor receptor assay with clinical parameters improves risk classification for relapse and survival in head-and-neck squamous cell carcinoma. Int J Radiat Oncol Biol Phys. 2011;81: 331-338.
- 14. Licitra L, Mesia R, Rivera F, et al. Evaluation of EGFR gene copy number as a predictive biomarker for the efficacy of cetuximab in combination with chemotherapy in the first-line treatment of recurrent and/or metastatic squamous cell carcinoma of the head and neck: EXTREME study. Ann Oncol. 2011;22: 1078-1087.
- 15. Peruzzi B, Bottaro DP. Targeting the c-Met signaling pathway in cancer. Clin Cancer Res. 2006;12: 3657-3660.
- 16. Mandal M, Myers JN, Lippman SM, et al. Epithelial to mesenchymal transition in head and neck squamous carcinoma: association of Src activation with E-cadherin down-regulation, vimentin expression, and aggressive tumor features. Cancer. 2008;112: 2088-2100.
- 17. Basu D, Nguyen TT, Montone KT, et al. Evidence for mesenchymal-like sub-populations within squamous cell carcinomas possessing chemoresistance and phenotypic plasticity. Oncogene. 2010;29: 4170-4182.
- 18. Knowles LM, Stabile LP, Egloff AM, et al. HGF and c-Met participate in paracrine tumorigenic pathways in head and neck squamous cell cancer. Clin Cancer Res. 2009;15: 3740-3750.

- 19. Seiwert TY, Jagadeeswaran R, Faoro L, et al. The MET receptor tyrosine kinase is a potential novel therapeutic target for head and neck squamous cell carcinoma. Cancer Res. 2009;69: 3021-3031.
- 20. Ghadjar P, Blank-Liss W, Simcock M, et al. MET Y1253D-activating point mutation and development of distant metastasis in advanced head and neck cancers. Clin Exp Metastasis. 2009;26: 809-815.
- 21. Stransky N, Egloff AM, Tward AD, et al. The mutational landscape of head and neck squamous cell carcinoma. Science. 2011;333: 1157-1160.
- 22. Agrawal N, Frederick MJ, Pickering CR, et al. Exome Sequencing of Head and Neck Squamous Cell Carcinoma Reveals Inactivating Mutations in NOTCH1. Science. 2011;333: 1154-1157.
- 23. Xu H, Stabile LP, Gubish CT, Gooding WE, Grandis JR, Siegfried JM. Dual blockade of EGFR and c-Met abrogates redundant signaling and proliferation in head and neck carcinoma cells. Clin Cancer Res. 2011;17: 4425-4438.
- 24. Wilson TR, Fridlyand J, Yan Y, et al. Widespread potential for growth-factor-driven resistance to anticancer kinase inhibitors. Nature. 2012;487: 505-509.
- 25. Takahashi N, Yamada Y, Furuta K, et al. Serum levels of hepatocyte growth factor and epiregulin are associated with the prognosis on anti-EGFR antibody treatment in KRAS wild-type metastatic colorectal cancer. Br J Cancer. 2014;110: 2716-2727.
- 26. Yamada T, Takeuchi S, Kita K, et al. Hepatocyte growth factor induces resistance to anti-epidermal growth factor receptor antibody in lung cancer. J Thorac Oncol. 2012;7: 272-280.
- 27. Tanaka H, Kimura T, Kudoh S, et al. Reaction of plasma hepatocyte growth factor levels in non-small cell lung cancer patients treated with EGFR-TKIs. Int J Cancer. 2011;129: 1410-1416.
- 28. Baselga J, Trigo JM, Bourhis J, et al. Phase II multicenter study of the antiepidermal growth factor receptor monoclonal antibody cetuximab in combination with platinum-based chemotherapy in patients with platinum-refractory metastatic and/or recurrent squamous cell carcinoma of the head and neck. J Clin Oncol. 2005;23: 5568-5577.
- 29. Shin DM, Donato NJ, Perez-Soler R, et al. Epidermal growth factor receptor-targeted therapy with C225 and cisplatin in patients with head and neck cancer. Clin Cancer Res. 2001;7: 1204-1213.
- 30. Tabernero J, Ciardiello F, Rivera F, et al. Cetuximab administered once every second week to patients with metastatic colorectal cancer: a two-part pharmacokinetic/pharmacodynamic phase I dose-escalation study. Ann Oncol. 2010;21: 1537-1545.
- 31. Tabernero J, Pfeiffer P, Cervantes A. Administration of cetuximab every 2 weeks in the treatment of metastatic colorectal cancer: an effective, more convenient alternative to weekly administration? Oncologist. 2008;13: 113-119.
- 32. Tabernero J, Cervantes A, Rivera F, et al. Pharmacogenomic and pharmacoproteomic studies of cetuximab in metastatic colorectal cancer: biomarker analysis of a phase I dose-escalation study. J Clin Oncol. 2010;28: 1181-1189.
- 33. Bossi P, Kornek G, Lanzetta G, et al. Safety and feasibility of every-other-week maintenance cetuximab after first-line chemotherapy in patients with recurrent or metastatic head and neck squamous cell cancer. Head Neck. 2012.
- 34. Leef G, Thomas SM. Molecular communication between tumor-associated fibroblasts and head and neck squamous cell carcinoma. Oral Oncol. 2013;49: 381-386.
- 35. Kumar D, Kandl C, Hamilton CD, et al. Mitigation of Tumor-Associated Fibroblast-Facilitated Head and Neck Cancer Progression With Anti-Hepatocyte Growth Factor Antibody Ficlatuzumab. JAMA Otolaryngol Head Neck Surg. 2015;141: 1133-1139.
- 36. Chung CH, Seeley EH, Roder H, et al. Detection of tumor epidermal growth factor receptor pathway dependence by serum mass spectrometry in cancer patients. Cancer Epidemiol Biomarkers Prev. 2010;19: 358-365.
- 37. Stransky N, Egloff AM, Tward AD, et al. The Mutational Landscape of Head and Neck Squamous Cell Carcinoma. Science. 2011.

- 38. Zhao D, Wang SH, Feng Y, Hua CG, Zhao J, Tang XF. Intratumoral c-Met expression is associated with vascular endothelial growth factor C expression, lymphangiogenesis, and lymph node metastasis in oral squamous cell carcinoma: implications for use as a prognostic marker. Hum Pathol. 2011;42: 1514-1523. 39. Kuss I, Hathaway B, Ferris RL, Gooding W, Whiteside TL. Decreased absolute counts of T lymphocyte subsets and their relation to disease in squamous cell carcinoma of the head and neck. Clin Cancer Res. 2004;10: 3755-3762.
- 40. Dasgupta S, Bhattacharya-Chatterjee M, O'Malley BW, Jr., Chatterjee SK. Inhibition of NK cell activity through TGF-beta 1 by down-regulation of NKG2D in a murine model of head and neck cancer. J Immunol. 2005;175: 5541-5550.
- 41. Bauernhofer T, Kuss I, Henderson B, Baum AS, Whiteside TL. Preferential apoptosis of CD56dim natural killer cell subset in patients with cancer. Eur J Immunol. 2003;33: 119-124.
- 42. Ferris R, TL Whiteside, and S. Ferrone Clinical significance of downregulated antigen processing machinery in head and neck cancer. Clinical Cancer Research. 2006: in press.
- 43. Lopez-Albaitero A, Nayak JV, Ogino T, et al. Role of antigen-processing machinery in the in vitro resistance of squamous cell carcinoma of the head and neck cells to recognition by CTL. J Immunol. 2006;176: 3402-3409.
- 44. Singhal E, Sen P. Hepatocyte growth factor-induced c-Src-phosphatidylinositol 3-kinase-AKT-mammalian target of rapamycin pathway inhibits dendritic cell activation by blocking IkappaB kinase activity. Int J Biochem Cell Biol. 2011;43: 1134-1146.
- 45. Singhal E, Kumar P, Sen P. A novel role for Bruton's tyrosine kinase in hepatocyte growth factor-mediated immunoregulation of dendritic cells. J Biol Chem. 2011;286: 32054-32063.
- 46. List MA, D'Antonio LL, Cella DF, et al. The Performance Status Scale for Head and Neck Cancer Patients and the Functional Assessment of Cancer Therapy-Head and Neck Scale. A study of utility and validity. Cancer. 1996;77: 2294-2301.
- 47. Burtness B, Anadkat M, Basti S, et al. NCCN Task Force Report: Management of dermatologic and other toxicities associated with EGFR inhibition in patients with cancer. J Natl Compr Canc Netw. 2009;7 Suppl 1: S5-21; quiz S22-24.
- 48. Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009;45: 228-247.
- 49. Vermorken JB, Herbst RS, Leon X, Amellal N, Baselga J. Overview of the efficacy of cetuximab in recurrent and/or metastatic squamous cell carcinoma of the head and neck in patients who previously failed platinum-based therapies. Cancer. 2008;112: 2710-2719.
- 50. Machiels JP, Haddad RI, Fayette J, et al. Afatinib versus methotrexate as second-line treatment in patients with recurrent or metastatic squamous-cell carcinoma of the head and neck progressing on or after platinum-based therapy (LUX-Head & Neck 1): an open-label, randomised phase 3 trial. Lancet Oncol. 2015;16: 583-594.
- 51. Benjamini Y, Hochbert Y. Controlling the false discovery rate: a practical and powerful approach to multiple testing. J Royal Stat Society Series B. 2005;57: 290-300.
- 52. Lee JJ, Liu DD. A predictive probability design for phase II cancer clinical trials. Clin Trials. 2008;5: 93-106.